CLINICAL TRIAL: NCT02525874
Title: An Open-Label Study to Assess the Effects of BG00012 on Lymphocyte Subsets in Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: Effect of BG00012 on Lymphocyte Subsets and Immunoglobulins in Subjects With Relapsing Remitting Multiple Sclerosis (RRMS).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109MS310; 2015-001973-42 (EudraCT Number)
Record Dates: First submitted 2015-07-10; First posted 2015-08-18 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis
Keywords: Tecfidera; DMF; dimethyl fumarate
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dimethyl fumarate (Experimental): 120 mg twice daily (BID) for the first 7 days and 240 mg BID thereafter
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — Initial oral dose for 7 days with maintenance dose thereafter
  Other Names: BG00012; Tecfidera; DMF

SUMMARY:
The primary objective of the study is to evaluate the effect of BG00012 on lymphocyte subset counts during the first year of treatment in subjects with relapsing-remitting multiple sclerosis (RRMS). A secondary objective is to evaluate the pharmacodynamic effect on absolute lymphocyte counts (ALCs) and immunoglobulins (Igs) during the first year of treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects of childbearing potential (including female subjects who are post-menopausal for less than 1 year) must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment.
* Must have a confirmed diagnosis of RRMS according to the revised McDonald criteria (2010) [Polman 2011]

Key Exclusion Criteria:

* History of or positive test result at Screening for:
* human immunodeficiency virus
* hepatitis C virus antibody
* hepatitis B infection
* Drug or alcohol abuse within 1 year prior to Screening.
* Prior treatment with any of the following:
* cladribine
* mitoxantrone
* total lymphoid irradiation
* alemtuzumab
* T-cell or T-cell receptor vaccination
* any therapeutic monoclonal antibody, with the exception of natalizumab or daclizumab
* Treatment with any of the following medications or procedures within 6 months prior to Baseline (Day 1):
* DMF (given as Fumaderm®) or BG00012; enrollment will be limited to no more than 40 subjects (out of 200) with prior DMF exposure
* cyclosporine
* azathioprine
* methotrexate
* mycophenolate mofetil
* intravenous (IV) Ig
* plasmapheresis or cytapheresis

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2015-08-11 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2018-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (30):
- United States (14):
  - Research Site, Gilbert, Arizona
  - Research Site, Long Beach, California
  - Research Site, Ocala, Florida
  - Research Site, Oldsmar, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Overland Park, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Traverse City, Michigan
  - Research Site, Raleigh, North Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Tacoma, Washington
- Belgium (3):
  - Research Site, La Louvière, Hainaut
  - Research Site, Bruges, West-Vlaanderen
  - Research Site, Brasschaat
- Bulgaria (3):
  - Research Site, Plaven
  - Research Site, Pleven
  - Research Site, Sofia
- Research Site, Kuwait City, Kuwait
- Lithuania (3):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Vilnius
- Poland (5):
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Plewiska
  - Research Site, Szczecin
- Research Site, Umuttepe, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Derived] Mao-Draayer Y, Bar-Or A, Balashov K, Foley J, Smoot K, Longbrake EE, Robertson D, Mendoza JP, Lewin JB, Everage N, Bozin I, Lyons J, Mokliatchouk O, Bame E, Giuliani F. Real-World Safety and Effectiveness of Dimethyl Fumarate in Patients with MS: Results from the ESTEEM Phase 4 and PROCLAIM Phase 3 Studies with a Focus on Older Patients. Adv Ther. 2025 Jan;42(1):395-412. doi: 10.1007/s12325-024-03047-w. Epub 2024 Nov 21. PMID 39570545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 11 August 2015 to 23 April 2018 in Belgium, Bulgaria, Lithuania, Kuwait, Poland and United States.
Pre-assignment Details: A total of 218 participants were enrolled in the study of which 158 participants completed the study
Groups:
- Dimethyl Fumarate (BG00012): Participants received 120 mg BID orally for the first 7 days and 240 mg BID thereafter until 96 weeks.
Period: Overall Study
Arm/Group | Dimethyl Fumarate (BG00012)
Started | 218
Completed | 158
Not Completed | 60
Not completed — Other | 1
Not completed — Investigator Decision | 1
Not completed — Consent withdrawn | 22
Not completed — Non-compliance with study drug | 3
Not completed — Adverse Event | 17
Not completed — Lost to Follow-up | 7
Not completed — Disease progression, defined by protocol | 2
Not completed — Disease relapse | 4
Not completed — Alternative Treatment for MS | 2
Not completed — New lesions in Brain | 1

BASELINE CHARACTERISTICS:
Population: The pharmacodynamic (PD) population was defined as all participants who received at least 1 dose of study treatment and had at least 1 pharmacodynamic measurement after baseline.
Arm/Group | Dimethyl Fumarate (BG00012)
Number analyzed (Participants) | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 66
  Unknown or Not Reported | 146
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 60
  More than one race | 3
  Unknown or Not Reported | 145

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lymphocyte Subsets Counts up to 48 Weeks: T Cell, B Cell, Natural Killer Cell (TBNK)
Description: Lymphocyte subsets include T cell, B cell and Natural killer (NK) cells.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36 and Week 48
Population: The PD population was defined as all participants who received at least 1 dose of study treatment and had at least 1 pharmacodynamic measurement after baseline. Here 'Number analyzed' signifies number of participants analyzed at specified timepoint for each subset.
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter (cells/mm^3)
Groups:
- Dimethyl Fumarate (BG00012): Participants received 120 mg BID for the first 7 days and 240 mg BID thereafter until 96 weeks.
Arm/Group | Dimethyl Fumarate (BG00012)
Number analyzed (Participants) | 218
cells per cubic millimeter (cells/mm^3)
  B Cells: Baseline: number analyzed (Participants) | 216
  B Cells: Baseline | 235.9 (168.88)
  B Cells: Change at Week 4: number analyzed (Participants) | 209
  B Cells: Change at Week 4 | -18.8 (89.71)
  B Cells: Change at Week 8: number analyzed (Participants) | 206
  B Cells: Change at Week 8 | -48.2 (122.20)
  B Cells: Change at Week 12: number analyzed (Participants) | 209
  B Cells: Change at Week 12 | -65.9 (128.53)
  B Cells: Change at Week 24: number analyzed (Participants) | 206
  B Cells: Change at Week 24 | -76.5 (140.33)
  B Cells: Change at Week 36: number analyzed (Participants) | 195
  B Cells: Change at Week 36 | -70.1 (104.80)
  B Cells: Change at Week 48: number analyzed (Participants) | 193
  B Cells: Change at Week 48 | -60.7 (115.26)
  NK Cells: Baseline: number analyzed (Participants) | 216
  NK Cells: Baseline | 184.2 (107.12)
  NK Cells: Change at Week 4: number analyzed (Participants) | 209
  NK Cells: Change at Week 4 | 6.1 (84.66)
  NK Cells: Change at Week 8: number analyzed (Participants) | 206
  NK Cells: Change at Week 8 | -9.0 (89.55)
  NK Cells: Change at Week 12: number analyzed (Participants) | 209
  NK Cells: Change at Week 12 | -21.7 (90.82)
  NK Cells: Change at Week 24: number analyzed (Participants) | 206
  NK Cells: Change at Week 24 | -26.9 (88.06)
  NK Cells: Change at Week 36: number analyzed (Participants) | 195
  NK Cells: Change at Week 36 | -41.5 (90.37)
  NK Cells: Change at Week 48: number analyzed (Participants) | 193
  NK Cells: Change at Week 48 | -42.0 (104.88)
  T Cells: Baseline: number analyzed (Participants) | 216
  T Cells: Baseline | 1318.1 (544.00)
  T Cells: Change at Week 4: number analyzed (Participants) | 209
  T Cells: Change at Week 4 | -44.8 (383.55)
  T Cells: Change at Week 8: number analyzed (Participants) | 206
  T Cells: Change at Week 8 | -167.0 (482.86)
  T Cells: Change at Week 12: number analyzed (Participants) | 209
  T Cells: Change at Week 12 | -284.3 (527.58)
  T Cells: Change at Week 24: number analyzed (Participants) | 206
  T Cells: Change at Week 24 | -446.7 (542.06)
  T Cells: Change at Week 36: number analyzed (Participants) | 195
  T Cells: Change at Week 36 | -545.5 (550.87)
  T Cells: Change at Week 48: number analyzed (Participants) | 193
  T Cells: Change at Week 48 | -580.2 (551.52)
  CD4+ T cells: Baseline: number analyzed (Participants) | 216
  CD4+ T cells: Baseline | 879.0 (400.71)
  CD4+ T cells: Change at Week 4: number analyzed (Participants) | 209
  CD4+ T cells: Change at Week 4 | -27.4 (256.21)
  CD4+ T cells: Change at Week 8: number analyzed (Participants) | 206
  CD4+ T cells: Change at Week 8 | -95.4 (318.07)
  CD4+ T cells: Change at Week 12: number analyzed (Participants) | 209
  CD4+ T cells: Change at Week 12 | -176.8 (353.52)
  CD4+ T cells: Change at Week 24: number analyzed (Participants) | 206
  CD4+ T cells: Change at Week 24 | -269.8 (360.92)
  CD4+ T cells: Change at Week 36: number analyzed (Participants) | 195
  CD4+ T cells: Change at Week 36 | -329.7 (374.66)
  CD4+ T cells: Change at Week 48: number analyzed (Participants) | 193
  CD4+ T cells: Change at Week 48 | -352.6 (380.77)
  CD8+ T cells: Baseline: number analyzed (Participants) | 216
  CD8+ T cells: Baseline | 419.5 (203.76)
  CD8+ T cells:Change at Week 4: number analyzed (Participants) | 209
  CD8+ T cells:Change at Week 4 | -14.2 (147.21)
  CD8+ T cells:Change at Week 8: number analyzed (Participants) | 206
  CD8+ T cells:Change at Week 8 | -65.3 (181.65)
  CD8+ T cells:Change at Week 12: number analyzed (Participants) | 209
  CD8+ T cells:Change at Week 12 | -100.4 (193.28)
  CD8+ T cells:Change at Week 24: number analyzed (Participants) | 206
  CD8+ T cells:Change at Week 24 | -170.2 (201.14)
  CD8+ T cells:Change at Week 36: number analyzed (Participants) | 195
  CD8+ T cells:Change at Week 36 | -201.4 (203.10)
  CD8+ T cells:Change at Week 48: number analyzed (Participants) | 193
  CD8+ T cells:Change at Week 48 | -214.9 (203.62)

2. Primary Outcome: Change From Baseline in Lymphocyte Subsets Counts up to 48 Weeks: T-Cells Subsets
Description: T-cells subsets includes Activated CD4+ T-cell, Activated CD8+ T-cell, Activated CD8+ T-cell [CD38+], Activated Th (T helper) 1 phenotype, Activated Th17 phenotype, Activated Th2-enriched phenotype, Activated CD4+ T-cell [CD38+HLA-DR+], Activated CD4+ T-cell [HLA-DR+], Activated CD8+ T-cell [HLA-DR+], Central Memory (CM) CD4+ T-cell [CD45RA-CCR7+], CM CD4+ T-cell [CD45RA-CCR7+], CM CD8+ T-cell [CD45RA-CCR7+], Effector CD4+ T-cell [CD45RA+CCR7-], Effector CD8+ T-cell [CD45RA+CCR7-], Effector Memory (EM) CD4+ T-cell [CD45RA-CCR7-], EM CD8+ T-cell [CD45RA-CCR7-], Effector Regulatory T-cells, Effector CD4+ T-cell [CD45RA+CCR7-], Effector CD8+ T-cell [CD45RA+CCR7-], Naïve CD4+ T-cell [CD45RA+], Naïve CD8+ T-cell [CD45RA+], Naïve (N) CD8+ T-cell [CD45RA+], Naïve Regulatory T-cells, Terminal Effector Regulatory T-cells, Th1 phenotype, Th17 phenotype, Th2-enriched phenotype. Here, Change at week is represented as CW.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Dimethyl Fumarate (BG00012)
Number analyzed (Participants) | 218
cells/mm^3
  Activated CD4+ T-cell [CD38+]: Baseline: number analyzed (Participants) | 140
  Activated CD4+ T-cell [CD38+]: Baseline | 632.6 (305.86)
  Activated CD4+ T-cell [CD38+]: Change at Week 4: number analyzed (Participants) | 136
  Activated CD4+ T-cell [CD38+]: Change at Week 4 | 15.2 (241.73)
  Activated CD4+ T-cell [CD38+]: Change at Week 8: number analyzed (Participants) | 133
  Activated CD4+ T-cell [CD38+]: Change at Week 8 | -26.5 (241.47)
  Activated CD4+ T-cell [CD38+]: Change at Week 12: number analyzed (Participants) | 137
  Activated CD4+ T-cell [CD38+]: Change at Week 12 | -53.4 (246.22)
  Activated CD4+ T-cell [CD38+]: Change at Week 24: number analyzed (Participants) | 137
  Activated CD4+ T-cell [CD38+]: Change at Week 24 | -100.4 (263.58)
  Activated CD4+ T-cell [CD38+]: Change at Week 36: number analyzed (Participants) | 129
  Activated CD4+ T-cell [CD38+]: Change at Week 36 | -106.8 (308.03)
  Activated CD4+ T-cell [CD38+]: Change at Week 48: number analyzed (Participants) | 128
  Activated CD4+ T-cell [CD38+]: Change at Week 48 | -125.9 (273.26)
  Activated CD8+ T-cell ([CD38+HLA-DR+]): Baseline: number analyzed (Participants) | 216
  Activated CD8+ T-cell ([CD38+HLA-DR+]): Baseline | 22.9 (25.64)
  ActivatedCD8+T-cell(CD38+HLA-DR+):CW 4: number analyzed (Participants) | 208
  ActivatedCD8+T-cell(CD38+HLA-DR+):CW 4 | 3.9 (21.83)
  ActivatedCD8+T-cell(CD38+HLA-DR+):CW 8: number analyzed (Participants) | 206
  ActivatedCD8+T-cell(CD38+HLA-DR+):CW 8 | -2.2 (24.46)
  ActivatedCD8+T-cell(CD38+HLA-DR+):CW 12: number analyzed (Participants) | 208
  ActivatedCD8+T-cell(CD38+HLA-DR+):CW 12 | -3.4 (23.53)
  ActivatedCD8+T-cell(CD38+HLA-DR+):CW 24: number analyzed (Participants) | 206
  ActivatedCD8+T-cell(CD38+HLA-DR+):CW 24 | -5.8 (24.72)
  ActivatedCD8+T-cell(CD38+HLA-DR+):CW 36: number analyzed (Participants) | 195
  ActivatedCD8+T-cell(CD38+HLA-DR+):CW 36 | -7.9 (27.32)
  ActivatedCD8+T-cell(CD38+HLA-DR+):CW 48: number analyzed (Participants) | 193
  ActivatedCD8+T-cell(CD38+HLA-DR+):CW 48 | -7.7 (24.92)
  Activated CD8+ T-cell [CD38+]: Baseline: number analyzed (Participants) | 140
  Activated CD8+ T-cell [CD38+]: Baseline | 275.4 (158.04)
  Activated CD8+ T-cell [CD38+]: Change at Week 4: number analyzed (Participants) | 136
  Activated CD8+ T-cell [CD38+]: Change at Week 4 | 18.2 (118.67)
  Activated CD8+ T-cell [CD38+]: Change at Week 8: number analyzed (Participants) | 133
  Activated CD8+ T-cell [CD38+]: Change at Week 8 | -21.7 (126.38)
  Activated CD8+ T-cell [CD38+]: Change at Week 12: number analyzed (Participants) | 137
  Activated CD8+ T-cell [CD38+]: Change at Week 12 | -50.8 (132.08)
  Activated CD8+ T-cell [CD38+]: Change at Week 24: number analyzed (Participants) | 137
  Activated CD8+ T-cell [CD38+]: Change at Week 24 | -91.8 (142.99)
  Activated CD8+ T-cell [CD38+]: Change at Week 36: number analyzed (Participants) | 129
  Activated CD8+ T-cell [CD38+]: Change at Week 36 | -99.3 (162.79)
  Activated CD8+ T-cell [CD38+]: Change at Week 48: number analyzed (Participants) | 128
  Activated CD8+ T-cell [CD38+]: Change at Week 48 | -114.3 (152.39)
  Activated Th1 phenotype: Baseline: number analyzed (Participants) | 216
  Activated Th1 phenotype: Baseline | 10.4 (6.52)
  Activated Th1 phenotype: Change at Week 4: number analyzed (Participants) | 208
  Activated Th1 phenotype: Change at Week 4 | 0.6 (6.09)
  Activated Th1 phenotype: Change at Week 8: number analyzed (Participants) | 206
  Activated Th1 phenotype: Change at Week 8 | -1.2 (6.87)
  Activated Th1 phenotype: Change at Week 12: number analyzed (Participants) | 209
  Activated Th1 phenotype: Change at Week 12 | -2.1 (6.63)
  Activated Th1 phenotype: Change at Week 24: number analyzed (Participants) | 206
  Activated Th1 phenotype: Change at Week 24 | -3.5 (6.47)
  Activated Th1 phenotype: Change at Week 36: number analyzed (Participants) | 195
  Activated Th1 phenotype: Change at Week 36 | -3.8 (6.82)
  Activated Th1 phenotype: Change at Week 48: number analyzed (Participants) | 193
  Activated Th1 phenotype: Change at Week 48 | -4.0 (6.50)
  Activated Th17 phenotype: Baseline: number analyzed (Participants) | 216
  Activated Th17 phenotype: Baseline | 1.1 (1.33)
  Activated Th17 phenotype: Change at Week 4: number analyzed (Participants) | 208
  Activated Th17 phenotype: Change at Week 4 | 0.0 (1.01)
  Activated Th17 phenotype: Change at Week 8: number analyzed (Participants) | 206
  Activated Th17 phenotype: Change at Week 8 | -0.2 (1.50)
  Activated Th17 phenotype: Change at Week 12: number analyzed (Participants) | 209
  Activated Th17 phenotype: Change at Week 12 | 0.0 (1.36)
  Activated Th17 phenotype: Change at Week 24: number analyzed (Participants) | 206
  Activated Th17 phenotype: Change at Week 24 | -0.4 (1.33)
  Activated Th17 phenotype: Change at Week 36: number analyzed (Participants) | 195
  Activated Th17 phenotype: Change at Week 36 | -0.4 (0.96)
  Activated Th17 phenotype: Change at Week 48: number analyzed (Participants) | 193
  Activated Th17 phenotype: Change at Week 48 | -0.3 (1.06)
  Activated Th2-enriched phenotype: Baseline: number analyzed (Participants) | 216
  Activated Th2-enriched phenotype: Baseline | 4.8 (4.83)
  Activated Th2-enriched phenotype: Change at Week 4: number analyzed (Participants) | 208
  Activated Th2-enriched phenotype: Change at Week 4 | 1.2 (5.36)
  Activated Th2-enriched phenotype: Change at Week 8: number analyzed (Participants) | 206
  Activated Th2-enriched phenotype: Change at Week 8 | 0.4 (6.13)
  Activated Th2-enriched phenotype: CW 12: number analyzed (Participants) | 209
  Activated Th2-enriched phenotype: CW 12 | 0.5 (6.54)
  Activated Th2-enriched phenotype: CW 24: number analyzed (Participants) | 206
  Activated Th2-enriched phenotype: CW 24 | 0.6 (6.84)
  Activated Th2-enriched phenotype: CW 36: number analyzed (Participants) | 195
  Activated Th2-enriched phenotype: CW 36 | 0.3 (6.57)
  Activated Th2-enriched phenotype: CW 48: number analyzed (Participants) | 193
  Activated Th2-enriched phenotype: CW 48 | 0.2 (5.14)
  Activated CD4+ T-cell [CD38+HLA-DR+]: Baseline: number analyzed (Participants) | 216
  Activated CD4+ T-cell [CD38+HLA-DR+]: Baseline | 17.3 (12.77)
  ActivatedCD4+ T-cell[CD38+HLA-DR+]:CW 4: number analyzed (Participants) | 208
  ActivatedCD4+ T-cell[CD38+HLA-DR+]:CW 4 | 2.5 (11.63)
  ActivatedCD4+ T-cell[CD38+HLA-DR+]:CW 8: number analyzed (Participants) | 206
  ActivatedCD4+ T-cell[CD38+HLA-DR+]:CW 8 | -0.3 (12.81)
  ActivatedCD4+ T-cell[CD38+HLA-DR+]:CW 12: number analyzed (Participants) | 209
  ActivatedCD4+ T-cell[CD38+HLA-DR+]:CW 12 | -1.6 (12.10)
  ActivatedCD4+ T-cell[CD38+HLA-DR+]:CW 24: number analyzed (Participants) | 206
  ActivatedCD4+ T-cell[CD38+HLA-DR+]:CW 24 | -3.2 (13.54)
  ActivatedCD4+ T-cell[CD38+HLA-DR+]:CW 36: number analyzed (Participants) | 195
  ActivatedCD4+ T-cell[CD38+HLA-DR+]:CW 36 | -4.1 (12.07)
  ActivatedCD4+ T-cell[CD38+HLA-DR+]:CW 48: number analyzed (Participants) | 193
  ActivatedCD4+ T-cell[CD38+HLA-DR+]:CW 48 | -4.2 (11.62)
  Activated CD4+ T-cell [HLA-DR+]: Baseline: number analyzed (Participants) | 140
  Activated CD4+ T-cell [HLA-DR+]: Baseline | 64.6 (32.45)
  Activated CD4+ T-cell [HLA-DR+]: Change at Week 4: number analyzed (Participants) | 136
  Activated CD4+ T-cell [HLA-DR+]: Change at Week 4 | 1.4 (27.95)
  Activated CD4+ T-cell [HLA-DR+]: Change at Week 8: number analyzed (Participants) | 133
  Activated CD4+ T-cell [HLA-DR+]: Change at Week 8 | -5.1 (38.57)
  Activated CD4+ T-cell [HLA-DR+]: Change at Week 12: number analyzed (Participants) | 137
  Activated CD4+ T-cell [HLA-DR+]: Change at Week 12 | -11.7 (31.71)
  Activated CD4+ T-cell [HLA-DR+]: Change at Week 24: number analyzed (Participants) | 137
  Activated CD4+ T-cell [HLA-DR+]: Change at Week 24 | -26.0 (30.09)
  Activated CD4+ T-cell [HLA-DR+]: Change at Week 36: number analyzed (Participants) | 129
  Activated CD4+ T-cell [HLA-DR+]: Change at Week 36 | -33.6 (36.39)
  Activated CD4+ T-cell [HLA-DR+]: Change at Week 48: number analyzed (Participants) | 128
  Activated CD4+ T-cell [HLA-DR+]: Change at Week 48 | -30.1 (38.57)
  Activated CD8+ T-cell [HLA-DR+]: Baseline: number analyzed (Participants) | 140
  Activated CD8+ T-cell [HLA-DR+]: Baseline | 81.2 (63.34)
  Activated CD8+ T-cell [HLA-DR+]: Change at Week 4: number analyzed (Participants) | 136
  Activated CD8+ T-cell [HLA-DR+]: Change at Week 4 | 2.5 (46.91)
  Activated CD8+ T-cell [HLA-DR+]: Change at Week 8: number analyzed (Participants) | 133
  Activated CD8+ T-cell [HLA-DR+]: Change at Week 8 | -5.5 (67.56)
  Activated CD8+ T-cell [HLA-DR+]: Change at Week 12: number analyzed (Participants) | 137
  Activated CD8+ T-cell [HLA-DR+]: Change at Week 12 | -18.2 (59.58)
  Activated CD8+ T-cell [HLA-DR+]: Change at Week 24: number analyzed (Participants) | 137
  Activated CD8+ T-cell [HLA-DR+]: Change at Week 24 | -38.1 (57.42)
  Activated CD8+ T-cell [HLA-DR+]: Change at Week 36: number analyzed (Participants) | 129
  Activated CD8+ T-cell [HLA-DR+]: Change at Week 36 | -48.3 (63.85)
  Activated CD8+ T-cell [HLA-DR+]: Change at Week 48: number analyzed (Participants) | 128
  Activated CD8+ T-cell [HLA-DR+]: Change at Week 48 | -49.3 (59.85)
  CM CD4+ T-cell [CD45RA-CCR7+]: Baseline: number analyzed (Participants) | 216
  CM CD4+ T-cell [CD45RA-CCR7+]: Baseline | 433.4 (220.05)
  CM CD4+ T-cell[CD45RA-CCR7+]:CW 4: number analyzed (Participants) | 208
  CM CD4+ T-cell[CD45RA-CCR7+]:CW 4 | -21.0 (185.07)
  CM CD4+ T-cell[CD45RA-CCR7+]:CW 8: number analyzed (Participants) | 206
  CM CD4+ T-cell[CD45RA-CCR7+]:CW 8 | -68.0 (196.02)
  CM CD4+T-cell[CD45RA-CCR7+]:CW 12: number analyzed (Participants) | 210
  CM CD4+T-cell[CD45RA-CCR7+]:CW 12 | -105.3 (206.11)
  CM CD4+T-cell[CD45RA-CCR7+]:CW 24: number analyzed (Participants) | 206
  CM CD4+T-cell[CD45RA-CCR7+]:CW 24 | -204.2 (220.61)
  CentralMemoryCD4+T-cell[CD45RA-CCR7+]:CW 36: number analyzed (Participants) | 195
  CentralMemoryCD4+T-cell[CD45RA-CCR7+]:CW 36 | -235.7 (221.44)
  CM CD4+T-cell[CD45RA-CCR7+]:CW 48: number analyzed (Participants) | 193
  CM CD4+T-cell[CD45RA-CCR7+]:CW 48 | -231.1 (225.25)
  CM CD8+ T-cell [CD45RA-CCR7+]: Baseline: number analyzed (Participants) | 216
  CM CD8+ T-cell [CD45RA-CCR7+]: Baseline | 59.9 (60.38)
  CM CD8+T-cell[CD45RA-CCR7+]:CW 4: number analyzed (Participants) | 208
  CM CD8+T-cell[CD45RA-CCR7+]:CW 4 | -9.6 (45.92)
  CM CD8+T-cell[CD45RA-CCR7+]:CW 8: number analyzed (Participants) | 206
  CM CD8+T-cell[CD45RA-CCR7+]:CW 8 | -16.9 (41.72)
  CM CD8+T-cell[CD45RA-CCR7+]:CW 12: number analyzed (Participants) | 209
  CM CD8+T-cell[CD45RA-CCR7+]:CW 12 | -22.0 (48.10)
  CM CD8+T-cell[CD45RA-CCR7+]:CW 24: number analyzed (Participants) | 206
  CM CD8+T-cell[CD45RA-CCR7+]:CW 24 | -39.2 (50.00)
  CM CD8+T-cell[CD45RA-CCR7+]:CW 36: number analyzed (Participants) | 195
  CM CD8+T-cell[CD45RA-CCR7+]:CW 36 | -44.3 (55.66)
  CM CD8+T-cell[CD45RA-CCR7+]:CW 48: number analyzed (Participants) | 193
  CM CD8+T-cell[CD45RA-CCR7+]:CW 48 | -45.9 (53.78)
  Effector CD4+ T-cell [CD45RA+CCR7-]: Baseline: number analyzed (Participants) | 216
  Effector CD4+ T-cell [CD45RA+CCR7-]: Baseline | 12.0 (23.21)
  Effector CD4+ T-cell[CD45RA+CCR7-]:Change atWeek4: number analyzed (Participants) | 208
  Effector CD4+ T-cell[CD45RA+CCR7-]:Change atWeek4 | 0.8 (12.66)
  Effector CD4+ T-cell[CD45RA+CCR7-]:Change atWeek8: number analyzed (Participants) | 206
  Effector CD4+ T-cell[CD45RA+CCR7-]:Change atWeek8 | -0.1 (12.58)
  Effector CD4+ T-cell[CD45RA+CCR7-]:Change atWeek12: number analyzed (Participants) | 210
  Effector CD4+ T-cell[CD45RA+CCR7-]:Change atWeek12 | -1.0 (12.43)
  Effector CD4+ T-cell[CD45RA+CCR7-]:CW 24: number analyzed (Participants) | 206
  Effector CD4+ T-cell[CD45RA+CCR7-]:CW 24 | -1.6 (17.42)
  Effector CD4+ T-cell[CD45RA+CCR7-]:CW 36: number analyzed (Participants) | 195
  Effector CD4+ T-cell[CD45RA+CCR7-]:CW 36 | -1.9 (19.20)
  Effector CD4+ T-cell[CD45RA+CCR7-]:CW 48: number analyzed (Participants) | 193
  Effector CD4+ T-cell[CD45RA+CCR7-]:CW 48 | -4.7 (18.75)
  Effector CD8+ T-cell [CD45RA+CCR7-]: Baseline: number analyzed (Participants) | 216
  Effector CD8+ T-cell [CD45RA+CCR7-]: Baseline | 101.4 (91.95)
  Effector CD8+ T-cell[CD45RA+CCR7-]:Change atWeek4: number analyzed (Participants) | 208
  Effector CD8+ T-cell[CD45RA+CCR7-]:Change atWeek4 | 1.7 (63.49)
  Effector CD8+ T-cell[CD45RA+CCR7-]:Change atWeek8: number analyzed (Participants) | 206
  Effector CD8+ T-cell[CD45RA+CCR7-]:Change atWeek8 | -15.9 (67.93)
  Effector CD8+ T-cell[CD45RA+CCR7-]:CW 12: number analyzed (Participants) | 209
  Effector CD8+ T-cell[CD45RA+CCR7-]:CW 12 | -15.2 (80.78)
  Effector CD8+ T-cell[CD45RA+CCR7-]:CW 24: number analyzed (Participants) | 206
  Effector CD8+ T-cell[CD45RA+CCR7-]:CW 24 | -42.8 (74.14)
  Effector CD8+ T-cell[CD45RA+CCR7-]:CW 36: number analyzed (Participants) | 195
  Effector CD8+ T-cell[CD45RA+CCR7-]:CW 36 | -55.6 (78.88)
  Effector CD8+ T-cell[CD45RA+CCR7-]:CW 48: number analyzed (Participants) | 193
  Effector CD8+ T-cell[CD45RA+CCR7-]:CW 48 | -50.9 (82.46)
  EM CD4+ T-cell [CD45RA-CCR7-]: Baseline: number analyzed (Participants) | 216
  EM CD4+ T-cell [CD45RA-CCR7-]: Baseline | 179.7 (86.21)
  EM CD4+ T-cell [CD45RA-CCR7-]: Change at Week 4: number analyzed (Participants) | 208
  EM CD4+ T-cell [CD45RA-CCR7-]: Change at Week 4 | 10.9 (87.56)
  EM CD4+ T-cell [CD45RA-CCR7-]: Change at Week 8: number analyzed (Participants) | 206
  EM CD4+ T-cell [CD45RA-CCR7-]: Change at Week 8 | -33.2 (88.53)
  EM CD4+ T-cell [CD45RA-CCR7-]: Change at Week 12: number analyzed (Participants) | 210
  EM CD4+ T-cell [CD45RA-CCR7-]: Change at Week 12 | -55.2 (90.59)
  EM CD4+ T-cell [CD45RA-CCR7-]: Change at Week 24: number analyzed (Participants) | 206
  EM CD4+ T-cell [CD45RA-CCR7-]: Change at Week 24 | -81.7 (106.78)
  EM CD4+ T-cell [CD45RA-CCR7-]: Change at Week 36: number analyzed (Participants) | 195
  EM CD4+ T-cell [CD45RA-CCR7-]: Change at Week 36 | -98.1 (111.77)
  EM CD4+ T-cell [CD45RA-CCR7-]: Change at Week 48: number analyzed (Participants) | 193
  EM CD4+ T-cell [CD45RA-CCR7-]: Change at Week 48 | -118.5 (100.25)
  EM CD8+ T-cell [CD45RA-CCR7-]: Baseline: number analyzed (Participants) | 216
  EM CD8+ T-cell [CD45RA-CCR7-]: Baseline | 129.0 (92.24)
  EM CD8+ T-cell [CD45RA-CCR7-]: Change at Week 4: number analyzed (Participants) | 208
  EM CD8+ T-cell [CD45RA-CCR7-]: Change at Week 4 | 7.6 (82.42)
  EM CD8+ T-cell [CD45RA-CCR7-]: Change at Week 8: number analyzed (Participants) | 206
  EM CD8+ T-cell [CD45RA-CCR7-]: Change at Week 8 | -22.8 (88.05)
  EM CD8+ T-cell [CD45RA-CCR7-]: Change at Week 12: number analyzed (Participants) | 209
  EM CD8+ T-cell [CD45RA-CCR7-]: Change at Week 12 | -41.0 (85.82)
  EM CD8+ T-cell [CD45RA-CCR7-]: Change at Week 24: number analyzed (Participants) | 206
  EM CD8+ T-cell [CD45RA-CCR7-]: Change at Week 24 | -69.9 (90.17)
  EM CD8+ T-cell [CD45RA-CCR7-]: Change at Week 36: number analyzed (Participants) | 195
  EM CD8+ T-cell [CD45RA-CCR7-]: Change at Week 36 | -80.3 (96.19)
  EM CD8+ T-cell [CD45RA-CCR7-]: Change at Week 48: number analyzed (Participants) | 193
  EM CD8+ T-cell [CD45RA-CCR7-]: Change at Week 48 | -90.3 (97.07)
  Effector Regulatory T-cells: Baseline: number analyzed (Participants) | 216
  Effector Regulatory T-cells: Baseline | 56.1 (28.88)
  Effector Regulatory T-cells: Change at Week 4: number analyzed (Participants) | 208
  Effector Regulatory T-cells: Change at Week 4 | 0.6 (26.13)
  Effector Regulatory T-cells: Change at Week 8: number analyzed (Participants) | 206
  Effector Regulatory T-cells: Change at Week 8 | -7.1 (27.32)
  Effector Regulatory T-cells: Change at Week 12: number analyzed (Participants) | 210
  Effector Regulatory T-cells: Change at Week 12 | -12.7 (25.81)
  Effector Regulatory T-cells: Change at Week 24: number analyzed (Participants) | 206
  Effector Regulatory T-cells: Change at Week 24 | -20.3 (28.31)
  Effector Regulatory T-cells: Change at Week 36: number analyzed (Participants) | 195
  Effector Regulatory T-cells: Change at Week 36 | -25.8 (31.50)
  Effector Regulatory T-cells: Change at Week 48: number analyzed (Participants) | 193
  Effector Regulatory T-cells: Change at Week 48 | -25.1 (29.73)
  Memory CD4+ T-cell [CD45RA-]: Baseline: number analyzed (Participants) | 216
  Memory CD4+ T-cell [CD45RA-]: Baseline | 617.7 (256.07)
  Memory CD4+ T-cell [CD45RA-]: Change at Week 4: number analyzed (Participants) | 208
  Memory CD4+ T-cell [CD45RA-]: Change at Week 4 | -6.2 (233.54)
  Memory CD4+ T-cell [CD45RA-]: Change at Week 8: number analyzed (Participants) | 206
  Memory CD4+ T-cell [CD45RA-]: Change at Week 8 | -100.9 (252.99)
  Memory CD4+ T-cell [CD45RA-]: Change at Week 12: number analyzed (Participants) | 210
  Memory CD4+ T-cell [CD45RA-]: Change at Week 12 | -157.7 (269.36)
  Memory CD4+ T-cell [CD45RA-]: Change at Week 24: number analyzed (Participants) | 206
  Memory CD4+ T-cell [CD45RA-]: Change at Week 24 | -287.7 (291.97)
  Memory CD4+ T-cell [CD45RA-]: Change at Week 36: number analyzed (Participants) | 195
  Memory CD4+ T-cell [CD45RA-]: Change at Week 36 | -335.0 (299.23)
  Memory CD4+ T-cell [CD45RA-]: Change at Week 48: number analyzed (Participants) | 193
  Memory CD4+ T-cell [CD45RA-]: Change at Week 48 | -349.9 (289.24)
  Memory CD8+ T-cell [CD45RA-]: Baseline: number analyzed (Participants) | 216
  Memory CD8+ T-cell [CD45RA-]: Baseline | 187.5 (126.58)
  Memory CD8+ T-cell [CD45RA-]: Change at Week 4: number analyzed (Participants) | 208
  Memory CD8+ T-cell [CD45RA-]: Change at Week 4 | -4.7 (97.59)
  Memory CD8+ T-cell [CD45RA-]: Change at Week 8: number analyzed (Participants) | 206
  Memory CD8+ T-cell [CD45RA-]: Change at Week 8 | -40.9 (109.49)
  Memory CD8+ T-cell [CD45RA-]: Change at Week 12: number analyzed (Participants) | 209
  Memory CD8+ T-cell [CD45RA-]: Change at Week 12 | -64.0 (118.89)
  Memory CD8+ T-cell [CD45RA-]: Change at Week 24: number analyzed (Participants) | 206
  Memory CD8+ T-cell [CD45RA-]: Change at Week 24 | -108.6 (119.94)
  Memory CD8+ T-cell [CD45RA-]: Change at Week 36: number analyzed (Participants) | 195
  Memory CD8+ T-cell [CD45RA-]: Change at Week 36 | -124.9 (126.30)
  Memory CD8+ T-cell [CD45RA-]: Change at Week 48: number analyzed (Participants) | 193
  Memory CD8+ T-cell [CD45RA-]: Change at Week 48 | -136.3 (129.68)
  Naïve CD4+ T-cell [CD45RA+CCR7+]: Baseline: number analyzed (Participants) | 216
  Naïve CD4+ T-cell [CD45RA+CCR7+]: Baseline | 400.9 (261.16)
  Naïve CD4+ T-cell [CD45RA+CCR7+]: Change at Week 4: number analyzed (Participants) | 208
  Naïve CD4+ T-cell [CD45RA+CCR7+]: Change at Week 4 | -10.5 (175.86)
  Naïve CD4+ T-cell [CD45RA+CCR7+]: Change at Week 8: number analyzed (Participants) | 206
  Naïve CD4+ T-cell [CD45RA+CCR7+]: Change at Week 8 | -16.4 (169.60)
  Naïve CD4+ T-cell[CD45RA+CCR7+]:Change at Week 12: number analyzed (Participants) | 210
  Naïve CD4+ T-cell[CD45RA+CCR7+]:Change at Week 12 | -11.8 (177.35)
  Naïve CD4+ T-cell[CD45RA+CCR7+]:Change at Week 24: number analyzed (Participants) | 206
  Naïve CD4+ T-cell[CD45RA+CCR7+]:Change at Week 24 | -31.7 (190.17)
  Naïve CD4+ T-cell[CD45RA+CCR7+]:Change at Week 36: number analyzed (Participants) | 195
  Naïve CD4+ T-cell[CD45RA+CCR7+]:Change at Week 36 | -29.3 (204.15)
  Naïve CD4+ T-cell[CD45RA+CCR7+]:Change at Week 48: number analyzed (Participants) | 193
  Naïve CD4+ T-cell[CD45RA+CCR7+]:Change at Week 48 | -34.4 (197.57)
  Naïve CD4+ T-cell [CD45RA+]: Baseline: number analyzed (Participants) | 216
  Naïve CD4+ T-cell [CD45RA+]: Baseline | 416.7 (268.35)
  Naïve CD4+ T-cell [CD45RA+]: Change at Week 4: number analyzed (Participants) | 208
  Naïve CD4+ T-cell [CD45RA+]: Change at Week 4 | -8.6 (177.59)
  Naïve CD4+ T-cell [CD45RA+]: Change at Week 8: number analyzed (Participants) | 206
  Naïve CD4+ T-cell [CD45RA+]: Change at Week 8 | -15.6 (173.25)
  Naïve CD4+ T-cell [CD45RA+]: Change at Week 12: number analyzed (Participants) | 210
  Naïve CD4+ T-cell [CD45RA+]: Change at Week 12 | -10.2 (185.67)
  Naïve CD4+ T-cell [CD45RA+]: Change at Week 24: number analyzed (Participants) | 206
  Naïve CD4+ T-cell [CD45RA+]: Change at Week 24 | -33.6 (193.78)
  Naïve CD4+ T-cell [CD45RA+]: Change at Week 36: number analyzed (Participants) | 195
  Naïve CD4+ T-cell [CD45RA+]: Change at Week 36 | -30.2 (214.46)
  Naïve CD4+ T-cell [CD45RA+]: Change at Week 48: number analyzed (Participants) | 193
  Naïve CD4+ T-cell [CD45RA+]: Change at Week 48 | -37.0 (206.10)
  Naïve CD8+ T-cell [CD45RA+CCR7+]: Baseline: number analyzed (Participants) | 216
  Naïve CD8+ T-cell [CD45RA+CCR7+]: Baseline | 160.1 (108.32)
  Naïve CD8+ T-cell [CD45RA+CCR7+]: Change at Week 4: number analyzed (Participants) | 208
  Naïve CD8+ T-cell [CD45RA+CCR7+]: Change at Week 4 | -11.6 (79.05)
  Naïve CD8+ T-cell [CD45RA+CCR7+]: Change at Week 8: number analyzed (Participants) | 206
  Naïve CD8+ T-cell [CD45RA+CCR7+]: Change at Week 8 | -12.4 (75.66)
  Naïve CD8+ T-cell[CD45RA+CCR7+]:Change at Week 12: number analyzed (Participants) | 209
  Naïve CD8+ T-cell[CD45RA+CCR7+]:Change at Week 12 | -22.0 (73.23)
  Naïve CD8+ T-cell[CD45RA+CCR7+]:Change at Week 24: number analyzed (Participants) | 206
  Naïve CD8+ T-cell[CD45RA+CCR7+]:Change at Week 24 | -41.3 (77.22)
  Naïve CD8+ T-cell[CD45RA+CCR7+]:Change at Week 36: number analyzed (Participants) | 195
  Naïve CD8+ T-cell[CD45RA+CCR7+]:Change at Week 36 | -49.0 (88.78)
  Naïve CD8+ T-cell[CD45RA+CCR7+]:Change at Week 48: number analyzed (Participants) | 193
  Naïve CD8+ T-cell[CD45RA+CCR7+]:Change at Week 48 | -50.9 (80.43)
  Naïve CD8+ T-cell [CD45RA+]: Baseline: number analyzed (Participants) | 216
  Naïve CD8+ T-cell [CD45RA+]: Baseline | 258.0 (150.73)
  Naïve CD8+ T-cell [CD45RA+]: Change at Week 4: number analyzed (Participants) | 208
  Naïve CD8+ T-cell [CD45RA+]: Change at Week 4 | -11.7 (118.68)
  Naïve CD8+ T-cell [CD45RA+]: Change at Week 8: number analyzed (Participants) | 206
  Naïve CD8+ T-cell [CD45RA+]: Change at Week 8 | -28.3 (118.33)
  Naïve CD8+ T-cell [CD45RA+]: Change at Week 12: number analyzed (Participants) | 209
  Naïve CD8+ T-cell [CD45RA+]: Change at Week 12 | -39.7 (131.27)
  Naïve CD8+ T-cell [CD45RA+]: Change at Week 24: number analyzed (Participants) | 206
  Naïve CD8+ T-cell [CD45RA+]: Change at Week 24 | -82.4 (134.00)
  Naïve CD8+ T-cell [CD45RA+]: Change at Week 36: number analyzed (Participants) | 195
  Naïve CD8+ T-cell [CD45RA+]: Change at Week 36 | -106.1 (139.47)
  Naïve CD8+ T-cell [CD45RA+]: Change at Week 48: number analyzed (Participants) | 193
  Naïve CD8+ T-cell [CD45RA+]: Change at Week 48 | -103.4 (138.84)
  Naïve Regulatory T-cells: Baseline: number analyzed (Participants) | 216
  Naïve Regulatory T-cells: Baseline | 15.8 (13.44)
  Naïve Regulatory T-cells: Change at Week 4: number analyzed (Participants) | 208
  Naïve Regulatory T-cells: Change at Week 4 | -0.1 (11.90)
  Naïve Regulatory T-cells: Change at Week 8: number analyzed (Participants) | 206
  Naïve Regulatory T-cells: Change at Week 8 | -0.4 (12.19)
  Naïve Regulatory T-cells: Change at Week 12: number analyzed (Participants) | 210
  Naïve Regulatory T-cells: Change at Week 12 | -0.7 (9.84)
  Naïve Regulatory T-cells: Change at Week 24: number analyzed (Participants) | 206
  Naïve Regulatory T-cells: Change at Week 24 | -0.4 (11.87)
  Naïve Regulatory T-cells: Change at Week 36: number analyzed (Participants) | 195
  Naïve Regulatory T-cells: Change at Week 36 | 0.1 (12.07)
  Naïve Regulatory T-cells: Change at Week 48: number analyzed (Participants) | 193
  Naïve Regulatory T-cells: Change at Week 48 | -0.1 (10.25)
  Regulatory T-cells: Baseline: number analyzed (Participants) | 216
  Regulatory T-cells: Baseline | 71.5 (36.60)
  Regulatory T-cells: Change at Week 4: number analyzed (Participants) | 208
  Regulatory T-cells: Change at Week 4 | 1.0 (34.31)
  Regulatory T-cells: Change at Week 8: number analyzed (Participants) | 206
  Regulatory T-cells: Change at Week 8 | -7.3 (35.01)
  Regulatory T-cells: Change at Week 12: number analyzed (Participants) | 210
  Regulatory T-cells: Change at Week 12 | -13.3 (32.12)
  Regulatory T-cells: Change at Week 24: number analyzed (Participants) | 206
  Regulatory T-cells: Change at Week 24 | -20.0 (36.77)
  Regulatory T-cells: Change at Week 36: number analyzed (Participants) | 195
  Regulatory T-cells: Change at Week 36 | -25.7 (40.18)
  Regulatory T-cells: Change at Week 48: number analyzed (Participants) | 193
  Regulatory T-cells: Change at Week 48 | -24.4 (36.09)
  Terminal Effector Regulatory T-cells: Baseline: number analyzed (Participants) | 140
  Terminal Effector Regulatory T-cells: Baseline | 327.2 (168.48)
  Terminal Effector Regulatory T-cells: CW 4: number analyzed (Participants) | 136
  Terminal Effector Regulatory T-cells: CW 4 | 16.6 (158.45)
  Terminal Effector Regulatory T-cells: CW 8: number analyzed (Participants) | 133
  Terminal Effector Regulatory T-cells: CW 8 | -4.4 (167.36)
  Terminal Effector Regulatory T-cells: CW 12: number analyzed (Participants) | 137
  Terminal Effector Regulatory T-cells: CW 12 | -17.6 (167.80)
  Terminal Effector Regulatory T-cells: CW 24: number analyzed (Participants) | 137
  Terminal Effector Regulatory T-cells: CW 24 | -58.3 (174.97)
  Terminal Effector Regulatory T-cells: CW 36: number analyzed (Participants) | 129
  Terminal Effector Regulatory T-cells: CW 36 | -97.2 (199.08)
  Terminal Effector Regulatory T-cells: CW 48: number analyzed (Participants) | 128
  Terminal Effector Regulatory T-cells: CW 48 | -98.6 (186.01)
  Th1 phenotype: Baseline: number analyzed (Participants) | 216
  Th1 phenotype: Baseline | 329.5 (153.17)
  Th1 phenotype: Change at Week 4: number analyzed (Participants) | 208
  Th1 phenotype: Change at Week 4 | -14.7 (127.21)
  Th1 phenotype: Change at Week 8: number analyzed (Participants) | 206
  Th1 phenotype: Change at Week 8 | -65.4 (147.25)
  Th1 phenotype: Change at Week 12: number analyzed (Participants) | 209
  Th1 phenotype: Change at Week 12 | -102.1 (149.63)
  Th1 phenotype: Change at Week 24: number analyzed (Participants) | 206
  Th1 phenotype: Change at Week 24 | -159.2 (172.24)
  Th1 phenotype: Change at Week 36: number analyzed (Participants) | 195
  Th1 phenotype: Change at Week 36 | -183.0 (177.40)
  Th1 phenotype: Change at Week 48: number analyzed (Participants) | 193
  Th1 phenotype: Change at Week 48 | -187.4 (172.19)
  Th17 phenotype: Baseline: number analyzed (Participants) | 216
  Th17 phenotype: Baseline | 61.9 (40.76)
  Th17 phenotype: Change at Week 4: number analyzed (Participants) | 208
  Th17 phenotype: Change at Week 4 | -0.5 (37.46)
  Th17 phenotype: Change at Week 8: number analyzed (Participants) | 206
  Th17 phenotype: Change at Week 8 | -7.3 (39.10)
  Th17 phenotype: Change at Week 12: number analyzed (Participants) | 209
  Th17 phenotype: Change at Week 12 | -1.1 (45.74)
  Th17 phenotype: Change at Week 24: number analyzed (Participants) | 206
  Th17 phenotype: Change at Week 24 | -24.6 (42.79)
  Th17 phenotype: Change at Week 36: number analyzed (Participants) | 195
  Th17 phenotype: Change at Week 36 | -35.1 (39.56)
  Th17 phenotype: Change at Week 48: number analyzed (Participants) | 193
  Th17 phenotype: Change at Week 48 | -30.1 (39.12)
  Th2-enriched phenotype: Baseline: number analyzed (Participants) | 216
  Th2-enriched phenotype: Baseline | 562.7 (289.42)
  Th2-enriched phenotype: Change at Week 4: number analyzed (Participants) | 208
  Th2-enriched phenotype: Change at Week 4 | -0.6 (211.18)
  Th2-enriched phenotype: Change at Week 8: number analyzed (Participants) | 206
  Th2-enriched phenotype: Change at Week 8 | -31.5 (227.69)
  Th2-enriched phenotype: Change at Week 12: number analyzed (Participants) | 209
  Th2-enriched phenotype: Change at Week 12 | -54.0 (210.95)
  Th2-enriched phenotype: Change at Week 24: number analyzed (Participants) | 206
  Th2-enriched phenotype: Change at Week 24 | -96.7 (241.83)
  Th2-enriched phenotype: Change at Week 36: number analyzed (Participants) | 195
  Th2-enriched phenotype: Change at Week 36 | -97.7 (267.45)
  Th2-enriched phenotype: Change at Week 48: number analyzed (Participants) | 193
  Th2-enriched phenotype: Change at Week 48 | -125.2 (242.46)

3. Primary Outcome: Change From Baseline in Lymphocyte Subsets Counts up to 48 Weeks: B-Cell Subsets
Description: B-cell subsets include CD10+ Transitional B cells, CD138+ Plasma Cells, Ig (Immunoglobulin) D+ Memory B cells [non-class switched], IgD- Memory B cells [class switched], Naïve B cells, Plasma Cells [CD10-], Transitional B-cells and Plasmablasts. Here, Change at week is represented as CW.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Dimethyl Fumarate (BG00012)
Number analyzed (Participants) | 218
cells/mm^3
  CD10+ Transitional B cells: Baseline: number analyzed (Participants) | 216
  CD10+ Transitional B cells: Baseline | 9.4 (9.93)
  CD10+ Transitional B cells: Change at Week 4: number analyzed (Participants) | 195
  CD10+ Transitional B cells: Change at Week 4 | -1.2 (7.98)
  CD10+ Transitional B cells: Change at Week 8: number analyzed (Participants) | 200
  CD10+ Transitional B cells: Change at Week 8 | -0.4 (8.73)
  CD10+ Transitional B cells: Change at Week 12: number analyzed (Participants) | 210
  CD10+ Transitional B cells: Change at Week 12 | -0.4 (9.09)
  CD10+ Transitional B cells: Change at Week 24: number analyzed (Participants) | 205
  CD10+ Transitional B cells: Change at Week 24 | 3.6 (10.16)
  CD10+ Transitional B cells: Change at Week 36: number analyzed (Participants) | 195
  CD10+ Transitional B cells: Change at Week 36 | 2.8 (9.53)
  CD10+ Transitional B cells: Change at Week 48: number analyzed (Participants) | 193
  CD10+ Transitional B cells: Change at Week 48 | 5.7 (13.53)
  CD138+ Plasma Cells: Baseline: number analyzed (Participants) | 216
  CD138+ Plasma Cells: Baseline | 0.26 (0.289)
  CD138+ Plasma Cells: Change at Week 4: number analyzed (Participants) | 195
  CD138+ Plasma Cells: Change at Week 4 | -0.02 (0.367)
  CD138+ Plasma Cells: Change at Week 8: number analyzed (Participants) | 200
  CD138+ Plasma Cells: Change at Week 8 | -0.12 (0.291)
  CD138+ Plasma Cells: Change at Week 12: number analyzed (Participants) | 210
  CD138+ Plasma Cells: Change at Week 12 | -0.15 (0.288)
  CD138+ Plasma Cells: Change at Week 24: number analyzed (Participants) | 205
  CD138+ Plasma Cells: Change at Week 24 | -0.21 (0.297)
  CD138+ Plasma Cells: Change at Week 36: number analyzed (Participants) | 195
  CD138+ Plasma Cells: Change at Week 36 | -0.21 (0.327)
  CD138+ Plasma Cells: Change at Week 48: number analyzed (Participants) | 193
  CD138+ Plasma Cells: Change at Week 48 | -0.19 (0.318)
  IgD+ Memory B cells [non-class switched]: Baseline: number analyzed (Participants) | 216
  IgD+ Memory B cells [non-class switched]: Baseline | 37.8 (36.96)
  IgD+ Memory B cells[non-class switched]: CW 4: number analyzed (Participants) | 195
  IgD+ Memory B cells[non-class switched]: CW 4 | -8.9 (26.18)
  IgD+ Memory B cells[non-class switched]: CW 8: number analyzed (Participants) | 200
  IgD+ Memory B cells[non-class switched]: CW 8 | -12.4 (29.27)
  IgD+ Memory B cells[non-class switched]: CW 12: number analyzed (Participants) | 210
  IgD+ Memory B cells[non-class switched]: CW 12 | -12.1 (29.13)
  IgD+ Memory B cells[non-class switched]: CW 24: number analyzed (Participants) | 205
  IgD+ Memory B cells[non-class switched]: CW 24 | -17.6 (31.39)
  IgD+ Memory B cells[non-class switched]: CW 36: number analyzed (Participants) | 195
  IgD+ Memory B cells[non-class switched]: CW 36 | -19.6 (31.61)
  IgD+ Memory B cells [non-class switched]: CW 48: number analyzed (Participants) | 193
  IgD+ Memory B cells [non-class switched]: CW 48 | -13.4 (34.89)
  IgD- Memory B cells [class switched]: Baseline: number analyzed (Participants) | 216
  IgD- Memory B cells [class switched]: Baseline | 50.4 (56.97)
  IgD- Memory B cells [class switched]: CW 4: number analyzed (Participants) | 195
  IgD- Memory B cells [class switched]: CW 4 | -8.7 (32.20)
  IgD- Memory B cells [class switched]: CW 8: number analyzed (Participants) | 200
  IgD- Memory B cells [class switched]: CW 8 | -17.7 (44.42)
  IgD- Memory B cells [class switched]: CW 12: number analyzed (Participants) | 210
  IgD- Memory B cells [class switched]: CW 12 | -23.1 (44.76)
  IgD- Memory B cells [class switched]: CW 24: number analyzed (Participants) | 205
  IgD- Memory B cells [class switched]: CW 24 | -29.5 (49.95)
  IgD- Memory B cells [class switched]: CW 36: number analyzed (Participants) | 195
  IgD- Memory B cells [class switched]: CW 36 | 49.95 (32.64)
  IgD- Memory B cells [class switched]: CW 48: number analyzed (Participants) | 193
  IgD- Memory B cells [class switched]: CW 48 | -27.4 (38.33)
  Naïve B cells: Baseline: number analyzed (Participants) | 216
  Naïve B cells: Baseline | 197.2 (140.48)
  Naïve B cells: Change at Week 4: number analyzed (Participants) | 195
  Naïve B cells: Change at Week 4 | -21.5 (82.43)
  Naïve B cells: Change at Week 8: number analyzed (Participants) | 200
  Naïve B cells: Change at Week 8 | -37.2 (95.32)
  Naïve B cells: Change at Week 12: number analyzed (Participants) | 210
  Naïve B cells: Change at Week 12 | -43.1 (99.72)
  Naïve B cells: Change at Week 24: number analyzed (Participants) | 205
  Naïve B cells: Change at Week 24 | -45.7 (114.46)
  Naïve B cells: Change at Week 36: number analyzed (Participants) | 195
  Naïve B cells: Change at Week 36 | -54.0 (94.94)
  Naïve B cells: Change at Week 48: number analyzed (Participants) | 193
  Naïve B cells: Change at Week 48 | -35.6 (107.79)
  Plasma Cells [CD10-]: Baseline: number analyzed (Participants) | 216
  Plasma Cells [CD10-]: Baseline | 0.63 (0.668)
  Plasma Cells [CD10-]: Change at Week 4: number analyzed (Participants) | 195
  Plasma Cells [CD10-]: Change at Week 4 | -0.02 (0.816)
  Plasma Cells [CD10-]: Change at Week 8: number analyzed (Participants) | 200
  Plasma Cells [CD10-]: Change at Week 8 | -0.11 (0.643)
  Plasma Cells [CD10-]: Change at Week 12: number analyzed (Participants) | 210
  Plasma Cells [CD10-]: Change at Week 12 | -0.18 (0.647)
  Plasma Cells [CD10-]: Change at Week 24: number analyzed (Participants) | 205
  Plasma Cells [CD10-]: Change at Week 24 | -0.34 (0.649)
  Plasma Cells [CD10-]: Change at Week 36: number analyzed (Participants) | 195
  Plasma Cells [CD10-]: Change at Week 36 | -0.33 (0.786)
  Plasma Cells [CD10-]: Change at Week 48: number analyzed (Participants) | 193
  Plasma Cells [CD10-]: Change at Week 48 | -0.38 (0.633)
  Transitional B-cells: Baseline: number analyzed (Participants) | 216
  Transitional B-cells: Baseline | 13.6 (13.61)
  Transitional B-cells: Change at Week 4: number analyzed (Participants) | 195
  Transitional B-cells: Change at Week 4 | -1.3 (11.44)
  Transitional B-cells: Change at Week 8: number analyzed (Participants) | 200
  Transitional B-cells: Change at Week 8 | 0.6 (12.97)
  Transitional B-cells: Change at Week 12: number analyzed (Participants) | 210
  Transitional B-cells: Change at Week 12 | 0.7 (13.41)
  Transitional B-cells: Change at Week 24: number analyzed (Participants) | 205
  Transitional B-cells: Change at Week 24 | 5.8 (15.60)
  Transitional B-cells: Change at Week 36: number analyzed (Participants) | 195
  Transitional B-cells: Change at Week 36 | 4.2 (13.20)
  Transitional B-cells: Change at Week 48: number analyzed (Participants) | 193
  Transitional B-cells: Change at Week 48 | 7.3 (18.56)
  Plasmablasts: Baseline: number analyzed (Participants) | 216
  Plasmablasts: Baseline | 0.91 (1.104)
  Plasmablasts: Change at Week 4: number analyzed (Participants) | 195
  Plasmablasts: Change at Week 4 | -0.04 (1.120)
  Plasmablasts: Change at Week 8: number analyzed (Participants) | 200
  Plasmablasts: Change at Week 8 | -0.21 (1.062)
  Plasmablasts: Change at Week 12: number analyzed (Participants) | 210
  Plasmablasts: Change at Week 12 | -0.31 (1.024)
  Plasmablasts: Change at Week 24: number analyzed (Participants) | 205
  Plasmablasts: Change at Week 24 | -0.46 (1.106)
  Plasmablasts: Change at Week 36: number analyzed (Participants) | 195
  Plasmablasts: Change at Week 36 | -0.46 (1.228)
  Plasmablasts: Change at Week 48: number analyzed (Participants) | 193
  Plasmablasts: Change at Week 48 | -0.50 (1.084)

4. Primary Outcome: Change From Baseline in Lymphocyte Subsets Counts up to 48 Weeks: Myeloid and Natural Killer (NK) Cells
Description: Myeloid and natural killer cell subsets include CD56Bright NK cells, CD56Dim NK cells, Classical Monocytes, Myeloid dendritic cells, Non-classical Monocytes, Plasmacytoid dendritic cells, Total dendritic cells and Total monocytes [CD14+].
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Dimethyl Fumarate (BG00012)
Number analyzed (Participants) | 218
cells/mm^3
  CD56Bright NK cells: Baseline: number analyzed (Participants) | 216
  CD56Bright NK cells: Baseline | 14.0 (8.94)
  CD56Bright NK cells: Change at Week 4: number analyzed (Participants) | 209
  CD56Bright NK cells: Change at Week 4 | 1.8 (6.40)
  CD56Bright NK cells: Change at Week 8: number analyzed (Participants) | 206
  CD56Bright NK cells: Change at Week 8 | 1.8 (7.07)
  CD56Bright NK cells: Change at Week 12: number analyzed (Participants) | 210
  CD56Bright NK cells: Change at Week 12 | 1.3 (7.26)
  CD56Bright NK cells: Change at Week 24: number analyzed (Participants) | 206
  CD56Bright NK cells: Change at Week 24 | 2.1 (8.57)
  CD56Bright NK cells: Change at Week 36: number analyzed (Participants) | 195
  CD56Bright NK cells: Change at Week 36 | 2.3 (9.73)
  CD56Bright NK cells: Change at Week 48: number analyzed (Participants) | 193
  CD56Bright NK cells: Change at Week 48 | 2.1 (8.55)
  CD56Dim NK cells: Baseline: number analyzed (Participants) | 216
  CD56Dim NK cells: Baseline | 192.9 (130.45)
  CD56Dim NK cells: Change at Week 4: number analyzed (Participants) | 209
  CD56Dim NK cells: Change at Week 4 | -2.0 (102.59)
  CD56Dim NK cells: Change at Week 8: number analyzed (Participants) | 206
  CD56Dim NK cells: Change at Week 8 | -17.2 (102.92)
  CD56Dim NK cells: Change at Week 12: number analyzed (Participants) | 210
  CD56Dim NK cells: Change at Week 12 | -31.4 (92.14)
  CD56Dim NK cells: Change at Week 24: number analyzed (Participants) | 206
  CD56Dim NK cells: Change at Week 24 | -50.7 (101.34)
  CD56Dim NK cells: Change at Week 36: number analyzed (Participants) | 195
  CD56Dim NK cells: Change at Week 36 | -61.1 (102.96)
  CD56Dim NK cells: Change at Week 48: number analyzed (Participants) | 193
  CD56Dim NK cells: Change at Week 48 | -68.5 (129.83)
  Classical Monocytes: Baseline: number analyzed (Participants) | 216
  Classical Monocytes: Baseline | 301.4 (153.48)
  Classical Monocytes: Change at Week 4: number analyzed (Participants) | 209
  Classical Monocytes: Change at Week 4 | 7.5 (182.11)
  Classical Monocytes: Change at Week 8: number analyzed (Participants) | 206
  Classical Monocytes: Change at Week 8 | 6.0 (165.07)
  Classical Monocytes: Change at Week 12: number analyzed (Participants) | 210
  Classical Monocytes: Change at Week 12 | 9.3 (197.84)
  Classical Monocytes: Change at Week 24: number analyzed (Participants) | 206
  Classical Monocytes: Change at Week 24 | -8.7 (151.23)
  Classical Monocytes: Change at Week 36: number analyzed (Participants) | 195
  Classical Monocytes: Change at Week 36 | -1.5 (163.62)
  Classical Monocytes: Change at Week 48: number analyzed (Participants) | 193
  Classical Monocytes: Change at Week 48 | -0.8 (153.24)
  Myeloid dendritic cells: Baseline: number analyzed (Participants) | 216
  Myeloid dendritic cells: Baseline | 24.96 (16.315)
  Myeloid dendritic cells: Change at Week 4: number analyzed (Participants) | 209
  Myeloid dendritic cells: Change at Week 4 | 1.46 (18.111)
  Myeloid dendritic cells: Change at Week 8: number analyzed (Participants) | 206
  Myeloid dendritic cells: Change at Week 8 | -0.61 (17.670)
  Myeloid dendritic cells: Change at Week 12: number analyzed (Participants) | 210
  Myeloid dendritic cells: Change at Week 12 | -0.23 (17.932)
  Myeloid dendritic cells: Change at Week 24: number analyzed (Participants) | 206
  Myeloid dendritic cells: Change at Week 24 | 3.02 (17.882)
  Myeloid dendritic cells: Change at Week 36: number analyzed (Participants) | 195
  Myeloid dendritic cells: Change at Week 36 | 3.63 (18.779)
  Myeloid dendritic cells: Change at Week 48: number analyzed (Participants) | 193
  Myeloid dendritic cells: Change at Week 48 | -6.20 (17.780)
  Non-classical Monocytes: Baseline: number analyzed (Participants) | 216
  Non-classical Monocytes: Baseline | 32.0 (22.88)
  Non-classical Monocytes: Change at Week 4: number analyzed (Participants) | 209
  Non-classical Monocytes: Change at Week 4 | 2.2 (29.82)
  Non-classical Monocytes: Change at Week 8: number analyzed (Participants) | 206
  Non-classical Monocytes: Change at Week 8 | -1.9 (30.14)
  Non-classical Monocytes: Change at Week 12: number analyzed (Participants) | 210
  Non-classical Monocytes: Change at Week 12 | -10.8 (23.82)
  Non-classical Monocytes: Change at Week 24: number analyzed (Participants) | 206
  Non-classical Monocytes: Change at Week 24 | -6.9 (27.65)
  Non-classical Monocytes: Change at Week 36: number analyzed (Participants) | 195
  Non-classical Monocytes: Change at Week 36 | -10.6 (24.24)
  Non-classical Monocytes: Change at Week 48: number analyzed (Participants) | 193
  Non-classical Monocytes: Change at Week 48 | -9.2 (24.37)
  Plasmacytoid dendritic cells: Baseline: number analyzed (Participants) | 216
  Plasmacytoid dendritic cells: Baseline | 6.52 (4.617)
  Plasmacytoid dendritic cells: Change at Week 4: number analyzed (Participants) | 209
  Plasmacytoid dendritic cells: Change at Week 4 | 0.00 (5.168)
  Plasmacytoid dendritic cells: Change at Week 8: number analyzed (Participants) | 206
  Plasmacytoid dendritic cells: Change at Week 8 | 0.30 (6.427)
  Plasmacytoid dendritic cells: Change at Week 12: number analyzed (Participants) | 210
  Plasmacytoid dendritic cells: Change at Week 12 | -0.86 (4.575)
  Plasmacytoid dendritic cells: Change at Week 24: number analyzed (Participants) | 206
  Plasmacytoid dendritic cells: Change at Week 24 | -0.69 (4.138)
  Plasmacytoid dendritic cells: Change at Week 36: number analyzed (Participants) | 195
  Plasmacytoid dendritic cells: Change at Week 36 | -0.80 (4.086)
  Plasmacytoid dendritic cells: Change at Week 48: number analyzed (Participants) | 193
  Plasmacytoid dendritic cells: Change at Week 48 | -2.22 (4.509)
  Total dendritic cells: Baseline: number analyzed (Participants) | 216
  Total dendritic cells: Baseline | 35.4 (19.92)
  Total dendritic cells: Change at Week 4: number analyzed (Participants) | 209
  Total dendritic cells: Change at Week 4 | 2.0 (22.35)
  Total dendritic cells: Change at Week 8: number analyzed (Participants) | 206
  Total dendritic cells: Change at Week 8 | -1.3 (21.68)
  Total dendritic cells: Change at Week 12: number analyzed (Participants) | 210
  Total dendritic cells: Change at Week 12 | -1.9 (21.07)
  Total dendritic cells: Change at Week 24: number analyzed (Participants) | 206
  Total dendritic cells: Change at Week 24 | 1.6 (21.89)
  Total dendritic cells: Change at Week 36: number analyzed (Participants) | 195
  Total dendritic cells: Change at Week 36 | 2.5 (22.19)
  Total dendritic cells: Change at Week 48: number analyzed (Participants) | 193
  Total dendritic cells: Change at Week 48 | -9.1 (22.77)
  Total monocytes [CD14+]: Baseline: number analyzed (Participants) | 216
  Total monocytes [CD14+]: Baseline | 374.6 (179.05)
  Total monocytes [CD14+]: Change at Week 4: number analyzed (Participants) | 209
  Total monocytes [CD14+]: Change at Week 4 | 26.9 (201.63)
  Total monocytes [CD14+]: Change at Week 8: number analyzed (Participants) | 206
  Total monocytes [CD14+]: Change at Week 8 | 12.6 (189.91)
  Total monocytes [CD14+]: Change at Week 12: number analyzed (Participants) | 210
  Total monocytes [CD14+]: Change at Week 12 | 14.4 (211.67)
  Total monocytes [CD14+]: Change at Week 24: number analyzed (Participants) | 206
  Total monocytes [CD14+]: Change at Week 24 | -19.3 (174.82)
  Total monocytes [CD14+]: Change at Week 36: number analyzed (Participants) | 195
  Total monocytes [CD14+]: Change at Week 36 | -21.7 (186.41)
  Total monocytes [CD14+]: Change at Week 48: number analyzed (Participants) | 193
  Total monocytes [CD14+]: Change at Week 48 | -19.2 (175.10)

5. Primary Outcome: Change From Baseline in Lymphocyte Subsets Counts up to 48 Weeks: T-Cell Cytokines
Description: T-cell cytokine subsets include IFN (interferon) g+ (% of CD4+ T cells), IFNg+ (% of CD8+ T cells), IFNg+ (% of memory CD4+ T cells), IFNg+ (% of memory CD8+ T cells), IL- (interleukin) 17A+/IFNg- (% of CD4+ T cells), IL-17A+/IFNg- (% of CD8+ T cells), IL-17A+/IFNg- (% of memory CD4+ T cells), IL-17A+/IFNg- (% of memory CD8+ T cells), IL-2+ (% of CD4+ T cells), IL-2+ (% of CD8+ T cells), IL-2+ (% of memory CD4+ T cells), IL-2+ (% of memory CD8+ T cells), IL-4+ (% of CD4+ T cells), IL-4+ (% of CD8+ T cells), IL-4+ (% of memory CD4+ T cells) and IL-4+ (% of memory CD8+ T cells). Here, Change at week is represented as CW.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Dimethyl Fumarate (BG00012)
Number analyzed (Participants) | 218
cells/mm^3
  IFNg+ (% of CD4+ T cells): Baseline: number analyzed (Participants) | 210
  IFNg+ (% of CD4+ T cells): Baseline | 3.340 (2.7365)
  IFNg+ (% of CD4+ T cells): Change at Week 4: number analyzed (Participants) | 193
  IFNg+ (% of CD4+ T cells): Change at Week 4 | 0.090 (2.2350)
  IFNg+ (% of CD4+ T cells): Change at Week 8: number analyzed (Participants) | 187
  IFNg+ (% of CD4+ T cells): Change at Week 8 | -0.356 (1.9676)
  IFNg+ (% of CD4+ T cells): Change at Week12: number analyzed (Participants) | 195
  IFNg+ (% of CD4+ T cells): Change at Week12 | -0.729 (2.1570)
  IFNg+ (% of CD4+ T cells): Change at Week24: number analyzed (Participants) | 193
  IFNg+ (% of CD4+ T cells): Change at Week24 | -1.134 (2.4239)
  IFNg+ (% of CD4+ T cells): Change at Week36: number analyzed (Participants) | 180
  IFNg+ (% of CD4+ T cells): Change at Week36 | -1.511 (2.5109)
  IFNg+ (% of CD4+ T cells): Change at Week48: number analyzed (Participants) | 182
  IFNg+ (% of CD4+ T cells): Change at Week48 | -1.222 (2.3513)
  IFNg+ (% of CD8+ T cells): Baseline: number analyzed (Participants) | 125
  IFNg+ (% of CD8+ T cells): Baseline | 6.166 (4.6199)
  IFNg+ (% of CD8+ T cells): Change at Week 4: number analyzed (Participants) | 118
  IFNg+ (% of CD8+ T cells): Change at Week 4 | 0.493 (2.8636)
  IFNg+ (% of CD8+ T cells): Change at Week 8: number analyzed (Participants) | 113
  IFNg+ (% of CD8+ T cells): Change at Week 8 | -0.264 (3.0735)
  IFNg+ (% of CD8+ T cells): Change at Week12: number analyzed (Participants) | 117
  IFNg+ (% of CD8+ T cells): Change at Week12 | -1.345 (3.3647)
  IFNg+ (% of CD8+ T cells): Change at Week24: number analyzed (Participants) | 118
  IFNg+ (% of CD8+ T cells): Change at Week24 | -1.650 (2.7202)
  IFNg+ (% of CD8+ T cells): Change at Week36: number analyzed (Participants) | 109
  IFNg+ (% of CD8+ T cells): Change at Week36 | -1.922 (4.1425)
  IFNg+ (% of CD8+ T cells): Change at Week48: number analyzed (Participants) | 111
  IFNg+ (% of CD8+ T cells): Change at Week48 | -1.306 (4.3931)
  IFNg+ (% of memory CD4+ T cells): Baseline: number analyzed (Participants) | 210
  IFNg+ (% of memory CD4+ T cells): Baseline | 4.518 (3.0417)
  IFNg+ (% of memory CD4+ T cells): CW 4: number analyzed (Participants) | 193
  IFNg+ (% of memory CD4+ T cells): CW 4 | 0.050 (2.5996)
  IFNg+ (% of memory CD4+ T cells): CW 8: number analyzed (Participants) | 187
  IFNg+ (% of memory CD4+ T cells): CW 8 | -0.295 (2.6287)
  IFNg+ (% of memory CD4+ T cells): CW 12: number analyzed (Participants) | 195
  IFNg+ (% of memory CD4+ T cells): CW 12 | -0.851 (2.8590)
  IFNg+ (% of memory CD4+ T cells): CW 24: number analyzed (Participants) | 193
  IFNg+ (% of memory CD4+ T cells): CW 24 | -1.019 (2.8120)
  IFNg+ (% of memory CD4+ T cells): CW 36: number analyzed (Participants) | 180
  IFNg+ (% of memory CD4+ T cells): CW 36 | -1.804 (2.6448)
  IFNg+ (% of memory CD4+ T cells): CW 48: number analyzed (Participants) | 182
  IFNg+ (% of memory CD4+ T cells): CW 48 | -1.369 (3.0958)
  IFNg+ (% of memory CD8+ T cells): Baseline: number analyzed (Participants) | 125
  IFNg+ (% of memory CD8+ T cells): Baseline | 8.795 (5.9060)
  IFNg+ (% of memory CD8+ T cells): CW 4: number analyzed (Participants) | 118
  IFNg+ (% of memory CD8+ T cells): CW 4 | 0.360 (3.6006)
  IFNg+ (% of memory CD8+ T cells): CW 8: number analyzed (Participants) | 113
  IFNg+ (% of memory CD8+ T cells): CW 8 | -0.285 (4.2645)
  IFNg+ (% of memory CD8+ T cells): CW 12: number analyzed (Participants) | 117
  IFNg+ (% of memory CD8+ T cells): CW 12 | -1.543 (3.7393)
  IFNg+ (% of memory CD8+ T cells): CW 24: number analyzed (Participants) | 118
  IFNg+ (% of memory CD8+ T cells): CW 24 | -0.964 (3.6799)
  IFNg+ (% of memory CD8+ T cells): CW 36: number analyzed (Participants) | 109
  IFNg+ (% of memory CD8+ T cells): CW 36 | -2.035 (5.3349)
  IFNg+ (% of memory CD8+ T cells): CW 48: number analyzed (Participants) | 111
  IFNg+ (% of memory CD8+ T cells): CW 48 | -0.497 (5.3126)
  IL-17A+/IFNg- (% of CD4+ T cells): Baseline: number analyzed (Participants) | 210
  IL-17A+/IFNg- (% of CD4+ T cells): Baseline | 1.244 (1.5863)
  IL-17A+/IFNg- (% of CD4+ T cells):Change at Week4: number analyzed (Participants) | 193
  IL-17A+/IFNg- (% of CD4+ T cells):Change at Week4 | 0.115 (1.9918)
  IL-17A+/IFNg- (% of CD4+ T cells):Change at Week8: number analyzed (Participants) | 187
  IL-17A+/IFNg- (% of CD4+ T cells):Change at Week8 | 0.131 (1.9097)
  IL-17A+/IFNg- (% of CD4+ T cells):Change at Week12: number analyzed (Participants) | 195
  IL-17A+/IFNg- (% of CD4+ T cells):Change at Week12 | 0.470 (2.3445)
  IL-17A+/IFNg- (% of CD4+ T cells):Change at Week24: number analyzed (Participants) | 193
  IL-17A+/IFNg- (% of CD4+ T cells):Change at Week24 | 0.165 (2.0104)
  IL-17A+/IFNg- (% of CD4+ T cells):Change at Week36: number analyzed (Participants) | 180
  IL-17A+/IFNg- (% of CD4+ T cells):Change at Week36 | 0.419 (2.5007)
  IL-17A+/IFNg- (% of CD4+ T cells):Change at Week48: number analyzed (Participants) | 182
  IL-17A+/IFNg- (% of CD4+ T cells):Change at Week48 | 1.693 (4.2412)
  IL-17A+/IFNg- (% of CD8+ T cells): Baseline: number analyzed (Participants) | 125
  IL-17A+/IFNg- (% of CD8+ T cells): Baseline | 0.455 (0.5309)
  IL-17A+/IFNg- (% of CD8+ T cells):Change at Week4: number analyzed (Participants) | 118
  IL-17A+/IFNg- (% of CD8+ T cells):Change at Week4 | 0.239 (1.3557)
  IL-17A+/IFNg- (% of CD8+ T cells):Change at Week8: number analyzed (Participants) | 113
  IL-17A+/IFNg- (% of CD8+ T cells):Change at Week8 | 0.032 (0.6448)
  IL-17A+/IFNg- (% of CD8+ T cells):Change at Week12: number analyzed (Participants) | 117
  IL-17A+/IFNg- (% of CD8+ T cells):Change at Week12 | 0.301 (0.8912)
  IL-17A+/IFNg- (% of CD8+ T cells):Change at Week24: number analyzed (Participants) | 118
  IL-17A+/IFNg- (% of CD8+ T cells):Change at Week24 | 0.289 (0.8526)
  IL-17A+/IFNg- (% of CD8+ T cells):Change at Week36: number analyzed (Participants) | 109
  IL-17A+/IFNg- (% of CD8+ T cells):Change at Week36 | 0.911 (1.3499)
  IL-17A+/IFNg- (% of CD8+ T cells):Change at Week48: number analyzed (Participants) | 111
  IL-17A+/IFNg- (% of CD8+ T cells):Change at Week48 | 1.457 (2.1499)
  IL-17A+/IFNg- (% of memory CD4+ T cells): Baseline: number analyzed (Participants) | 210
  IL-17A+/IFNg- (% of memory CD4+ T cells): Baseline | 1.075 (1.1770)
  IL-17A+/IFNg- (% of memory CD4+T cells): CW 4: number analyzed (Participants) | 193
  IL-17A+/IFNg- (% of memory CD4+T cells): CW 4 | 0.000 (1.3599)
  IL-17A+/IFNg- (% of memory CD4+T cells): CW 8: number analyzed (Participants) | 187
  IL-17A+/IFNg- (% of memory CD4+T cells): CW 8 | 0.040 (1.3593)
  IL-17A+/IFNg- (% of memory CD4+T cells): CW 12: number analyzed (Participants) | 195
  IL-17A+/IFNg- (% of memory CD4+T cells): CW 12 | 0.373 (1.7166)
  IL-17A+/IFNg- (% of memory CD4+T cells): CW 24: number analyzed (Participants) | 193
  IL-17A+/IFNg- (% of memory CD4+T cells): CW 24 | 0.228 (1.4980)
  IL-17A+/IFNg- (% of memory CD4+T cells): CW 36: number analyzed (Participants) | 180
  IL-17A+/IFNg- (% of memory CD4+T cells): CW 36 | 0.333 (1.8786)
  IL-17A+/IFNg- (% of memory CD4+T cells): CW 48: number analyzed (Participants) | 182
  IL-17A+/IFNg- (% of memory CD4+T cells): CW 48 | 1.255 (2.9557)
  IL-17A+/IFNg- (% of memory CD8+ T cells): Baseline: number analyzed (Participants) | 125
  IL-17A+/IFNg- (% of memory CD8+ T cells): Baseline | 0.155 (0.2356)
  IL-17A+/IFNg- (% of memory CD8+T cells): CW 4: number analyzed (Participants) | 118
  IL-17A+/IFNg- (% of memory CD8+T cells): CW 4 | 0.113 (0.6972)
  IL-17A+/IFNg- (% of memory CD8+T cells): CW 8: number analyzed (Participants) | 113
  IL-17A+/IFNg- (% of memory CD8+T cells): CW 8 | 0.027 (0.3641)
  IL-17A+/IFNg- (% of memory CD8+T cells): CW 12: number analyzed (Participants) | 117
  IL-17A+/IFNg- (% of memory CD8+T cells): CW 12 | 0.064 (0.3641)
  IL-17A+/IFNg- (% of memory CD8+T cells): CW 24: number analyzed (Participants) | 118
  IL-17A+/IFNg- (% of memory CD8+T cells): CW 24 | 0.254 (0.8682)
  IL-17A+/IFNg- (% of memory CD8+T cells): CW 36: number analyzed (Participants) | 109
  IL-17A+/IFNg- (% of memory CD8+T cells): CW 36 | 0.270 (0.6113)
  IL-17A+/IFNg- (% of memory CD8+T cells): CW 48: number analyzed (Participants) | 111
  IL-17A+/IFNg- (% of memory CD8+T cells): CW 48 | 0.680 (1.2842)
  IL-2+ (% of CD4+ T cells): Baseline: number analyzed (Participants) | 210
  IL-2+ (% of CD4+ T cells): Baseline | 5.177 (4.5225)
  IL-2+ (% of CD4+ T cells): Change at Week 4: number analyzed (Participants) | 193
  IL-2+ (% of CD4+ T cells): Change at Week 4 | 0.062 (3.4662)
  IL-2+ (% of CD4+ T cells): Change at Week 8: number analyzed (Participants) | 187
  IL-2+ (% of CD4+ T cells): Change at Week 8 | 0.149 (4.0713)
  IL-2+ (% of CD4+ T cells): Change at Week 12: number analyzed (Participants) | 195
  IL-2+ (% of CD4+ T cells): Change at Week 12 | -0.069 (4.0822)
  IL-2+ (% of CD4+ T cells): Change at Week 24: number analyzed (Participants) | 193
  IL-2+ (% of CD4+ T cells): Change at Week 24 | -0.448 (3.6280)
  IL-2+ (% of CD4+ T cells): Change at Week 36: number analyzed (Participants) | 180
  IL-2+ (% of CD4+ T cells): Change at Week 36 | -1.837 (3.8603)
  IL-2+ (% of CD4+ T cells): Change at Week 48: number analyzed (Participants) | 182
  IL-2+ (% of CD4+ T cells): Change at Week 48 | -1.840 (5.0951)
  IL-2+ (% of CD8+ T cells): Baseline: number analyzed (Participants) | 125
  IL-2+ (% of CD8+ T cells): Baseline | 1.180 (1.4533)
  IL-2+ (% of CD8+ T cells): Change at Week 4: number analyzed (Participants) | 118
  IL-2+ (% of CD8+ T cells): Change at Week 4 | -0.081 (1.2797)
  IL-2+ (% of CD8+ T cells): Change at Week 8: number analyzed (Participants) | 113
  IL-2+ (% of CD8+ T cells): Change at Week 8 | -0.227 (1.1579)
  IL-2+ (% of CD8+ T cells): Change at Week 12: number analyzed (Participants) | 117
  IL-2+ (% of CD8+ T cells): Change at Week 12 | -0.2622 (1.2601)
  IL-2+ (% of CD8+ T cells): Change at Week 24: number analyzed (Participants) | 118
  IL-2+ (% of CD8+ T cells): Change at Week 24 | -0.525 (1.0201)
  IL-2+ (% of CD8+ T cells): Change at Week 36: number analyzed (Participants) | 109
  IL-2+ (% of CD8+ T cells): Change at Week 36 | -0.547 (1.2886)
  IL-2+ (% of CD8+ T cells): Change at Week 48: number analyzed (Participants) | 111
  IL-2+ (% of CD8+ T cells): Change at Week 48 | -0.248 (1.1860)
  IL-2+ (% of memory CD4+ T cells): Baseline: number analyzed (Participants) | 210
  IL-2+ (% of memory CD4+ T cells): Baseline | 7.053 (5.6653)
  IL-2+ (% of memory CD4+ T cells): Change at Week 4: number analyzed (Participants) | 193
  IL-2+ (% of memory CD4+ T cells): Change at Week 4 | -0.105 (4.4131)
  IL-2+ (% of memory CD4+ T cells): Change at Week 8: number analyzed (Participants) | 187
  IL-2+ (% of memory CD4+ T cells): Change at Week 8 | 0.056 (4.6541)
  IL-2+ (% of memory CD4+ T cells): Change at Week12: number analyzed (Participants) | 195
  IL-2+ (% of memory CD4+ T cells): Change at Week12 | 0.012 (4.9241)
  IL-2+ (% of memory CD4+ T cells): Change at Week24: number analyzed (Participants) | 193
  IL-2+ (% of memory CD4+ T cells): Change at Week24 | 0.015 (4.6456)
  IL-2+ (% of memory CD4+ T cells): Change at Week36: number analyzed (Participants) | 180
  IL-2+ (% of memory CD4+ T cells): Change at Week36 | -2.140 (4.7723)
  IL-2+ (% of memory CD4+ T cells): Change at Week48: number analyzed (Participants) | 182
  IL-2+ (% of memory CD4+ T cells): Change at Week48 | -1.946 (5.6985)
  IL-2+ (% of memory CD8+ T cells): Baseline: number analyzed (Participants) | 125
  IL-2+ (% of memory CD8+ T cells): Baseline | 1.879 (1.7964)
  IL-2+ (% of memory CD8+ T cells): Change at Week 4: number analyzed (Participants) | 118
  IL-2+ (% of memory CD8+ T cells): Change at Week 4 | -0.218 (1.6838)
  IL-2+ (% of memory CD8+ T cells): Change at Week 8: number analyzed (Participants) | 113
  IL-2+ (% of memory CD8+ T cells): Change at Week 8 | -0.318 (1.7272)
  IL-2+ (% of memory CD8+ T cells): Change at Week12: number analyzed (Participants) | 117
  IL-2+ (% of memory CD8+ T cells): Change at Week12 | -0.115 (1.7354)
  IL-2+ (% of memory CD8+ T cells): Change at Week24: number analyzed (Participants) | 118
  IL-2+ (% of memory CD8+ T cells): Change at Week24 | -0.461 (1.4512)
  IL-2+ (% of memory CD8+ T cells): Change at Week36: number analyzed (Participants) | 109
  IL-2+ (% of memory CD8+ T cells): Change at Week36 | -0.803 (1.8525)
  IL-2+ (% of memory CD8+ T cells): Change at Week48: number analyzed (Participants) | 111
  IL-2+ (% of memory CD8+ T cells): Change at Week48 | -0.315 (2.0510)
  IL-4+ (% of CD4+ T cells: Baseline: number analyzed (Participants) | 210
  IL-4+ (% of CD4+ T cells: Baseline | 1.261 (1.1190)
  IL-4+ (% of CD4+ T cells): Change at Week 4: number analyzed (Participants) | 193
  IL-4+ (% of CD4+ T cells): Change at Week 4 | -0.150 (1.0429)
  IL-4+ (% of CD4+ T cells): Change at Week 8: number analyzed (Participants) | 187
  IL-4+ (% of CD4+ T cells): Change at Week 8 | -0.113 (1.2168)
  IL-4+ (% of CD4+ T cells): Change at Week12: number analyzed (Participants) | 195
  IL-4+ (% of CD4+ T cells): Change at Week12 | -0.370 (1.0594)
  IL-4+ (% of CD4+ T cells): Change at Week24: number analyzed (Participants) | 193
  IL-4+ (% of CD4+ T cells): Change at Week24 | -0.170 (1.1551)
  IL-4+ (% of CD4+ T cells): Change at Week36: number analyzed (Participants) | 180
  IL-4+ (% of CD4+ T cells): Change at Week36 | -0.376 (1.0920)
  IL-4+ (% of CD4+ T cells): Change at Week48: number analyzed (Participants) | 182
  IL-4+ (% of CD4+ T cells): Change at Week48 | 0.281 (4.7206)
  IL-4+ (% of CD8+ T cells): Baseline: number analyzed (Participants) | 125
  IL-4+ (% of CD8+ T cells): Baseline | 1.107 (1.2924)
  IL-4+ (% of CD8+ T cells): Change at Week 4: number analyzed (Participants) | 118
  IL-4+ (% of CD8+ T cells): Change at Week 4 | -0.222 (1.2163)
  IL-4+ (% of CD8+ T cells): Change at Week 8: number analyzed (Participants) | 113
  IL-4+ (% of CD8+ T cells): Change at Week 8 | -0.189 (1.3377)
  IL-4+ (% of CD8+ T cells): Change at Week12: number analyzed (Participants) | 117
  IL-4+ (% of CD8+ T cells): Change at Week12 | -0.553 (1.3754)
  IL-4+ (% of CD8+ T cells): Change at Week24: number analyzed (Participants) | 118
  IL-4+ (% of CD8+ T cells): Change at Week24 | -0.032 (1.3170)
  IL-4+ (% of CD8+ T cells): Change at Week36: number analyzed (Participants) | 109
  IL-4+ (% of CD8+ T cells): Change at Week36 | -0.195 (1.3334)
  IL-4+ (% of CD8+ T cells): Change at Week48: number analyzed (Participants) | 111
  IL-4+ (% of CD8+ T cells): Change at Week48 | 0.786 (1.3454)
  IL-4+ (% of memory CD4+ T cells): Baseline: number analyzed (Participants) | 210
  IL-4+ (% of memory CD4+ T cells): Baseline | 1.406 (1.2437)
  IL-4+ (% of memory CD4+ T cells): Change at Week 4: number analyzed (Participants) | 193
  IL-4+ (% of memory CD4+ T cells): Change at Week 4 | -0.128 (1.2649)
  IL-4+ (% of memory CD4+ T cells): Change at Week 8: number analyzed (Participants) | 187
  IL-4+ (% of memory CD4+ T cells): Change at Week 8 | -0.141 (1.4642)
  IL-4+ (% of memory CD4+ T cells): Change at Week12: number analyzed (Participants) | 195
  IL-4+ (% of memory CD4+ T cells): Change at Week12 | -0.412 (1.3656)
  IL-4+ (% of memory CD4+ T cells): Change at Week24: number analyzed (Participants) | 193
  IL-4+ (% of memory CD4+ T cells): Change at Week24 | -0.136 (1.3059)
  IL-4+ (% of memory CD4+ T cells): Change at Week36: number analyzed (Participants) | 180
  IL-4+ (% of memory CD4+ T cells): Change at Week36 | -0.266 (1.4005)
  IL-4+ (% of memory CD4+ T cells): Change at Week48: number analyzed (Participants) | 182
  IL-4+ (% of memory CD4+ T cells): Change at Week48 | 0.325 (1.7918)
  IL-4+ (% of memory CD8+ T cells): Baseline: number analyzed (Participants) | 125
  IL-4+ (% of memory CD8+ T cells): Baseline | 1.376 (1.8963)
  IL-4+ (% of memory CD8+ T cells): Change at Week 4: number analyzed (Participants) | 118
  IL-4+ (% of memory CD8+ T cells): Change at Week 4 | -0.180 (2.0821)
  IL-4+ (% of memory CD8+ T cells): Change at Week 8: number analyzed (Participants) | 113
  IL-4+ (% of memory CD8+ T cells): Change at Week 8 | -0.269 (1.9840)
  IL-4+ (% of memory CD8+ T cells): Change at Week12: number analyzed (Participants) | 117
  IL-4+ (% of memory CD8+ T cells): Change at Week12 | -0.795 (2.2486)
  IL-4+ (% of memory CD8+ T cells): Change at Week24: number analyzed (Participants) | 118
  IL-4+ (% of memory CD8+ T cells): Change at Week24 | 0.416 (2.3613)
  IL-4+ (% of memory CD8+ T cells): Change at Week36: number analyzed (Participants) | 109
  IL-4+ (% of memory CD8+ T cells): Change at Week36 | -0.284 (2.4433)
  IL-4+ (% of memory CD8+ T cells): Change at Week48: number analyzed (Participants) | 111
  IL-4+ (% of memory CD8+ T cells): Change at Week48 | 1.836 (2.7709)

6. Primary Outcome: Change From Baseline in Lymphocyte Subsets Counts up to 48 Weeks: Very Late Antigen-4 (VLA-4/Lymphocyte Function-Associated Antigen-1 (LFA-1) Antigen
Description: VLA-4/LFA-1 antigen subsets include CD11a+ (% of B cells), CD11a+ (% of T cells), CD11a+ (% of MNC), CD11a+ (% of dendritic cells [CD11c++]), CD11a+ (% of lymphocytes), CD11a+ (% of monocytes), CD11a+ (% of neutrophils), CD49d+ (% of B cells), CD49d+ (% of T cells), CD49d+ (% of MNC), CD49d+ (% of dendritic cells [CD11c++]), CD49d+ (% of lymphocytes), CD49d+ (% of monocytes) and CD49d+ (% of neutrophils).
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Dimethyl Fumarate (BG00012)
Number analyzed (Participants) | 218
cells/mm^3
  CD11a+ (% of B cells): Baseline: number analyzed (Participants) | 205
  CD11a+ (% of B cells): Baseline | 99.33 (2.106)
  CD11a+ (% of B cells): Change at Week 4: number analyzed (Participants) | 197
  CD11a+ (% of B cells): Change at Week 4 | 0.34 (2.497)
  CD11a+ (% of B cells): Change at Week 8: number analyzed (Participants) | 196
  CD11a+ (% of B cells): Change at Week 8 | 0.44 (2.203)
  CD11a+ (% of B cells): Change at Week 12: number analyzed (Participants) | 200
  CD11a+ (% of B cells): Change at Week 12 | 0.17 (2.534)
  CD11a+ (% of B cells): Change at Week 24: number analyzed (Participants) | 195
  CD11a+ (% of B cells): Change at Week 24 | 0.19 (2.549)
  CD11a+ (% of B cells): Change at Week 36: number analyzed (Participants) | 185
  CD11a+ (% of B cells): Change at Week 36 | -1.43 (11.406)
  CD11a+ (% of B cells): Change at Week 48: number analyzed (Participants) | 183
  CD11a+ (% of B cells): Change at Week 48 | -0.14 (7.751)
  CD11a+ (% of T cells): Baseline: number analyzed (Participants) | 205
  CD11a+ (% of T cells): Baseline | 99.90 (0.312)
  CD11a+ (% of T cells): Change at Week 4: number analyzed (Participants) | 197
  CD11a+ (% of T cells): Change at Week 4 | 0.05 (0.319)
  CD11a+ (% of T cells): Change at Week 8: number analyzed (Participants) | 196
  CD11a+ (% of T cells): Change at Week 8 | 0.07 (0.327)
  CD11a+ (% of T cells): Change at Week 12: number analyzed (Participants) | 200
  CD11a+ (% of T cells): Change at Week 12 | 0.06 (0.321)
  CD11a+ (% of T cells): Change at Week 24: number analyzed (Participants) | 195
  CD11a+ (% of T cells): Change at Week 24 | 0.02 (0.633)
  CD11a+ (% of T cells): Change at Week 36: number analyzed (Participants) | 185
  CD11a+ (% of T cells): Change at Week 36 | -1.29 (9.760)
  CD11a+ (% of T cells): Change at Week 48: number analyzed (Participants) | 183
  CD11a+ (% of T cells): Change at Week 48 | -0.53 (7.410)
  CD11a+ (% of MNC): Baseline: number analyzed (Participants) | 205
  CD11a+ (% of MNC): Baseline | 96.85 (3.089)
  CD11a+ (% of MNC): Change at Week 4: number analyzed (Participants) | 197
  CD11a+ (% of MNC): Change at Week 4 | 0.47 (3.630)
  CD11a+ (% of MNC): Change at Week 8: number analyzed (Participants) | 196
  CD11a+ (% of MNC): Change at Week 8 | 0.59 (3.532)
  CD11a+ (% of MNC): Change at Week 12: number analyzed (Participants) | 200
  CD11a+ (% of MNC): Change at Week 12 | 0.59 (3.710)
  CD11a+ (% of MNC): Change at Week 24: number analyzed (Participants) | 195
  CD11a+ (% of MNC): Change at Week 24 | -0.38 (3.963)
  CD11a+ (% of MNC): Change at Week 36: number analyzed (Participants) | 185
  CD11a+ (% of MNC): Change at Week 36 | -1.55 (10.918)
  CD11a+ (% of MNC): Change at Week 48: number analyzed (Participants) | 183
  CD11a+ (% of MNC): Change at Week 48 | -2.31 (8.402)
  CD11a+ (% of dendritic cells [CD11c++]): Baseline: number analyzed (Participants) | 205
  CD11a+ (% of dendritic cells [CD11c++]): Baseline | 99.81 (0.933)
  CD11a+ (% of dendritic cells [CD11c++]): CW 4: number analyzed (Participants) | 197
  CD11a+ (% of dendritic cells [CD11c++]): CW 4 | 0.04 (0.867)
  CD11a+ (% of dendritic cells [CD11c++]): CW 8: number analyzed (Participants) | 196
  CD11a+ (% of dendritic cells [CD11c++]): CW 8 | 0.02 (1.573)
  CD11a+ (% of dendritic cells [CD11c++]): CW 12: number analyzed (Participants) | 200
  CD11a+ (% of dendritic cells [CD11c++]): CW 12 | 0.10 (1.250)
  CD11a+ (% of dendritic cells [CD11c++]): CW 24: number analyzed (Participants) | 195
  CD11a+ (% of dendritic cells [CD11c++]): CW 24 | 0.01 (1.477)
  CD11a+ (% of dendritic cells [CD11c++]): CW 36: number analyzed (Participants) | 185
  CD11a+ (% of dendritic cells [CD11c++]): CW 36 | -1.27 (10.857)
  CD11a+ (% of dendritic cells [CD11c++]): CW 48: number analyzed (Participants) | 183
  CD11a+ (% of dendritic cells [CD11c++]): CW 48 | -0.84 (7.813)
  CD11a+ (% of lymphocytes): Baseline: number analyzed (Participants) | 205
  CD11a+ (% of lymphocytes): Baseline | 98.24 (1.870)
  CD11a+ (% of lymphocytes): Change at Week 4: number analyzed (Participants) | 197
  CD11a+ (% of lymphocytes): Change at Week 4 | 0.04 (2.227)
  CD11a+ (% of lymphocytes): Change at Week 8: number analyzed (Participants) | 196
  CD11a+ (% of lymphocytes): Change at Week 8 | 0.07 (2.649)
  CD11a+ (% of lymphocytes): Change at Week 12: number analyzed (Participants) | 200
  CD11a+ (% of lymphocytes): Change at Week 12 | 0.26 (2.604)
  CD11a+ (% of lymphocytes): Change at Week 24: number analyzed (Participants) | 195
  CD11a+ (% of lymphocytes): Change at Week 24 | -0.35 (2.519)
  CD11a+ (% of lymphocytes): Change at Week 36: number analyzed (Participants) | 185
  CD11a+ (% of lymphocytes): Change at Week 36 | -1.99 (10.532)
  CD11a+ (% of lymphocytes): Change at Week 48: number analyzed (Participants) | 183
  CD11a+ (% of lymphocytes): Change at Week 48 | -2.56 (8.696)
  CD11a+ (% of monocytes): Baseline: number analyzed (Participants) | 205
  CD11a+ (% of monocytes): Baseline | 98.00 (2.303)
  CD11a+ (% of monocytes): Change at Week 4: number analyzed (Participants) | 197
  CD11a+ (% of monocytes): Change at Week 4 | 0.29 (3.241)
  CD11a+ (% of monocytes): Change at Week 8: number analyzed (Participants) | 196
  CD11a+ (% of monocytes): Change at Week 8 | 0.92 (2.416)
  CD11a+ (% of monocytes): Change at Week 12: number analyzed (Participants) | 200
  CD11a+ (% of monocytes): Change at Week 12 | 0.77 (2.539)
  CD11a+ (% of monocytes): Change at Week 24: number analyzed (Participants) | 195
  CD11a+ (% of monocytes): Change at Week 24 | -0.40 (3.046)
  CD11a+ (% of monocytes): Change at Week 36: number analyzed (Participants) | 185
  CD11a+ (% of monocytes): Change at Week 36 | -0.36 (7.843)
  CD11a+ (% of monocytes): Change at Week 48: number analyzed (Participants) | 183
  CD11a+ (% of monocytes): Change at Week 48 | -1.52 (7.711)
  CD11a+ (% of neutrophils): Baseline: number analyzed (Participants) | 205
  CD11a+ (% of neutrophils): Baseline | 97.80 (5.352)
  CD11a+ (% of neutrophils): Change at Week 4: number analyzed (Participants) | 197
  CD11a+ (% of neutrophils): Change at Week 4 | 0.83 (6.672)
  CD11a+ (% of neutrophils): Change at Week 8: number analyzed (Participants) | 196
  CD11a+ (% of neutrophils): Change at Week 8 | 1.23 (5.675)
  CD11a+ (% of neutrophils): Change at Week 12: number analyzed (Participants) | 200
  CD11a+ (% of neutrophils): Change at Week 12 | 0.55 (6.113)
  CD11a+ (% of neutrophils): Change at Week 24: number analyzed (Participants) | 195
  CD11a+ (% of neutrophils): Change at Week 24 | 0.35 (9.220)
  CD11a+ (% of neutrophils): Change at Week 36: number analyzed (Participants) | 185
  CD11a+ (% of neutrophils): Change at Week 36 | -2.88 (18.513)
  CD11a+ (% of neutrophils): Change at Week 48: number analyzed (Participants) | 183
  CD11a+ (% of neutrophils): Change at Week 48 | 0.42 (10.736)
  CD49d+ (% of B cells): Baseline: number analyzed (Participants) | 205
  CD49d+ (% of B cells): Baseline | 99.87 (0.679)
  CD49d+ (% of B cells): Change at Week 4: number analyzed (Participants) | 197
  CD49d+ (% of B cells): Change at Week 4 | -0.50 (7.105)
  CD49d+ (% of B cells): Change at Week 8: number analyzed (Participants) | 196
  CD49d+ (% of B cells): Change at Week 8 | 0.00 (0.642)
  CD49d+ (% of B cells): Change at Week 12: number analyzed (Participants) | 200
  CD49d+ (% of B cells): Change at Week 12 | 0.01 (0.486)
  CD49d+ (% of B cells): Change at Week 24: number analyzed (Participants) | 194
  CD49d+ (% of B cells): Change at Week 24 | -0.01 (0.663)
  CD49d+ (% of B cells): Change at Week 36: number analyzed (Participants) | 185
  CD49d+ (% of B cells): Change at Week 36 | -0.07 (0.744)
  CD49d+ (% of B cells): Change at Week 48: number analyzed (Participants) | 183
  CD49d+ (% of B cells): Change at Week 48 | -0.04 (0.964)
  CD49d+ (% of T cells): Baseline: number analyzed (Participants) | 205
  CD49d+ (% of T cells): Baseline | 91.23 (4.427)
  CD49d+ (% of T cells): Change at Week 4: number analyzed (Participants) | 197
  CD49d+ (% of T cells): Change at Week 4 | -0.45 (6.909)
  CD49d+ (% of T cells): Change at Week 8: number analyzed (Participants) | 196
  CD49d+ (% of T cells): Change at Week 8 | -0.11 (2.055)
  CD49d+ (% of T cells): Change at Week 12: number analyzed (Participants) | 200
  CD49d+ (% of T cells): Change at Week 12 | -0.06 (1.930)
  CD49d+ (% of T cells): Change at Week 24: number analyzed (Participants) | 194
  CD49d+ (% of T cells): Change at Week 24 | -0.12 (2.209)
  CD49d+ (% of T cells): Change at Week 36: number analyzed (Participants) | 185
  CD49d+ (% of T cells): Change at Week 36 | -1.32 (4.256)
  CD49d+ (% of T cells): Change at Week 48: number analyzed (Participants) | 183
  CD49d+ (% of T cells): Change at Week 48 | -0.02 (2.935)
  CD49d+ (% of MNC): Baseline: number analyzed (Participants) | 205
  CD49d+ (% of MNC): Baseline | 86.79 (5.369)
  CD49d+ (% of MNC): Change at Week 4: number analyzed (Participants) | 197
  CD49d+ (% of MNC): Change at Week 4 | 0.23 (8.274)
  CD49d+ (% of MNC): Change at Week 8: number analyzed (Participants) | 196
  CD49d+ (% of MNC): Change at Week 8 | 0.38 (5.600)
  CD49d+ (% of MNC): Change at Week 12: number analyzed (Participants) | 200
  CD49d+ (% of MNC): Change at Week 12 | 0.85 (5.900)
  CD49d+ (% of MNC): Change at Week 24: number analyzed (Participants) | 194
  CD49d+ (% of MNC): Change at Week 24 | -0.07 (6.051)
  CD49d+ (% of MNC): Change at Week 36: number analyzed (Participants) | 185
  CD49d+ (% of MNC): Change at Week 36 | -0.46 (8.264)
  CD49d+ (% of MNC): Change at Week 48: number analyzed (Participants) | 183
  CD49d+ (% of MNC): Change at Week 48 | -1.25 (6.561)
  CD49d+ (% of dendritic cells [CD11c++]): Baseline: number analyzed (Participants) | 205
  CD49d+ (% of dendritic cells [CD11c++]): Baseline | 99.77 (0.771)
  CD49d+ (% of dendritic cells [CD11c++]): CW 4: number analyzed (Participants) | 197
  CD49d+ (% of dendritic cells [CD11c++]): CW 4 | -0.42 (7.185)
  CD49d+ (% of dendritic cells [CD11c++]): CW 8: number analyzed (Participants) | 196
  CD49d+ (% of dendritic cells [CD11c++]): CW 8 | 0.12 (0.874)
  CD49d+ (% of dendritic cells [CD11c++]): CW 12: number analyzed (Participants) | 200
  CD49d+ (% of dendritic cells [CD11c++]): CW 12 | 0.03 (1.252)
  CD49d+ (% of dendritic cells [CD11c++]): CW 24: number analyzed (Participants) | 194
  CD49d+ (% of dendritic cells [CD11c++]): CW 24 | 0.00 (1.162)
  CD49d+ (% of dendritic cells [CD11c++]): CW 36: number analyzed (Participants) | 185
  CD49d+ (% of dendritic cells [CD11c++]): CW 36 | -0.06 (1.532)
  CD49d+ (% of dendritic cells [CD11c++]): CW 48: number analyzed (Participants) | 183
  CD49d+ (% of dendritic cells [CD11c++]): CW 48 | -0.23 (1.530)
  CD49d+ (% of lymphocytes): Baseline: number analyzed (Participants) | 205
  CD49d+ (% of lymphocytes): Baseline | 91.29 (4.715)
  CD49d+ (% of lymphocytes): Change at Week 4: number analyzed (Participants) | 197
  CD49d+ (% of lymphocytes): Change at Week 4 | -0.31 (7.260)
  CD49d+ (% of lymphocytes): Change at Week 8: number analyzed (Participants) | 196
  CD49d+ (% of lymphocytes): Change at Week 8 | 0.03 (5.899)
  CD49d+ (% of lymphocytes): Change at Week 12: number analyzed (Participants) | 200
  CD49d+ (% of lymphocytes): Change at Week 12 | 0.44 (2.989)
  CD49d+ (% of lymphocytes): Change at Week 24: number analyzed (Participants) | 194
  CD49d+ (% of lymphocytes): Change at Week 24 | 0.01 (3.237)
  CD49d+ (% of lymphocytes): Change at Week 36: number analyzed (Participants) | 185
  CD49d+ (% of lymphocytes): Change at Week 36 | -0.75 (5.045)
  CD49d+ (% of lymphocytes): Change at Week 48: number analyzed (Participants) | 183
  CD49d+ (% of lymphocytes): Change at Week 48 | -1.10 (5.739)
  CD49d+ (% of monocytes): Baseline: number analyzed (Participants) | 205
  CD49d+ (% of monocytes): Baseline | 88.77 (8.126)
  CD49d+ (% of monocytes): Change at Week 4: number analyzed (Participants) | 197
  CD49d+ (% of monocytes): Change at Week 4 | 0.82 (10.895)
  CD49d+ (% of monocytes): Change at Week 8: number analyzed (Participants) | 196
  CD49d+ (% of monocytes): Change at Week 8 | 0.96 (10.161)
  CD49d+ (% of monocytes): Change at Week 12: number analyzed (Participants) | 200
  CD49d+ (% of monocytes): Change at Week 12 | 0.82 (10.350)
  CD49d+ (% of monocytes): Change at Week 24: number analyzed (Participants) | 194
  CD49d+ (% of monocytes): Change at Week 24 | 0.98 (9.793)
  CD49d+ (% of monocytes): Change at Week 36: number analyzed (Participants) | 185
  CD49d+ (% of monocytes): Change at Week 36 | 3.87 (9.683)
  CD49d+ (% of monocytes): Change at Week 48: number analyzed (Participants) | 183
  CD49d+ (% of monocytes): Change at Week 48 | 0.69 (10.594)
  CD49d+ (% of neutrophils): Baseline: number analyzed (Participants) | 205
  CD49d+ (% of neutrophils): Baseline | 5.61 (7.277)
  CD49d+ (% of neutrophils): Change at Week 4: number analyzed (Participants) | 197
  CD49d+ (% of neutrophils): Change at Week 4 | 4.43 (9.345)
  CD49d+ (% of neutrophils): Change at Week 8: number analyzed (Participants) | 196
  CD49d+ (% of neutrophils): Change at Week 8 | 1.17 (4.892)
  CD49d+ (% of neutrophils): Change at Week 12: number analyzed (Participants) | 200
  CD49d+ (% of neutrophils): Change at Week 12 | 0.27 (4.137)
  CD49d+ (% of neutrophils): Change at Week 24: number analyzed (Participants) | 194
  CD49d+ (% of neutrophils): Change at Week 24 | -0.67 (10.365)
  CD49d+ (% of neutrophils): Change at Week 36: number analyzed (Participants) | 185
  CD49d+ (% of neutrophils): Change at Week 36 | -0.29 (12.678)
  CD49d+ (% of neutrophils): Change at Week 48: number analyzed (Participants) | 183
  CD49d+ (% of neutrophils): Change at Week 48 | 0.92 (10.291)

7. Secondary Outcome: Change From Baseline in Immunoglobulin A (IgA) up to 48 Weeks
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36 and Week 48
Population: The PD population was defined as all participants who received at least 1 dose of study treatment and had at least 1 pharmacodynamic measurement after baseline. Here 'number analyzed' signifies number of participants analyzed at each timepoint.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Dimethyl Fumarate (BG00012)
Number analyzed (Participants) | 218
milligram per liter (mg/L)
  Baseline: number analyzed (Participants) | 216
  Baseline | 2116.5 (910.47)
  Change at Week 4: number analyzed (Participants) | 211
  Change at Week 4 | -120.0 (231.16)
  Change at Week 8: number analyzed (Participants) | 209
  Change at Week 8 | -112.8 (243.28)
  Change at Week 12: number analyzed (Participants) | 210
  Change at Week 12 | -93.6 (291.76)
  Change at Week 24: number analyzed (Participants) | 205
  Change at Week 24 | -101.5 (324.27)
  Change at Week 36: number analyzed (Participants) | 193
  Change at Week 36 | -65.1 (279.53)
  Change at Week 48: number analyzed (Participants) | 193
  Change at Week 48 | -94.9 (291.25)

8. Secondary Outcome: Change From Baseline in Immunoglobulin M (IgM) up to 48 Weeks
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Dimethyl Fumarate (BG00012)
Number analyzed (Participants) | 218
mg/L
  Baseline: number analyzed (Participants) | 216
  Baseline | 1330.1 (705.92)
  Change at Week 4: number analyzed (Participants) | 211
  Change at Week 4 | -68.9 (214.07)
  Change at Week 8: number analyzed (Participants) | 209
  Change at Week 8 | -23.2 (208.48)
  Change at Week 12: number analyzed (Participants) | 210
  Change at Week 12 | -18.8 (270.82)
  Change at Week 24: number analyzed (Participants) | 205
  Change at Week 24 | -36.9 (293.14)
  Change at Week 36: number analyzed (Participants) | 193
  Change at Week 36 | -19.4 (406.86)
  Change at Week 48: number analyzed (Participants) | 193
  Change at Week 48 | -96.8 (236.48)

9. Secondary Outcome: Change From Baseline in Immunoglobulin G (IgG) up to 48 Weeks
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Dimethyl Fumarate (BG00012)
Number analyzed (Participants) | 218
g/L
  Baseline: number analyzed (Participants) | 216
  Baseline | 10.51 (2.328)
  Change at Week 4: number analyzed (Participants) | 211
  Change at Week 4 | -0.77 (1.039)
  Change at Week 8: number analyzed (Participants) | 209
  Change at Week 8 | -0.64 (1.077)
  Change at Week 12: number analyzed (Participants) | 210
  Change at Week 12 | -0.44 (1.187)
  Change at Week 24: number analyzed (Participants) | 205
  Change at Week 24 | -0.62 (1.324)
  Change at Week 36: number analyzed (Participants) | 193
  Change at Week 36 | -0.36 (1.025)
  Change at Week 48: number analyzed (Participants) | 193
  Change at Week 48 | -0.53 (1.142)

10. Secondary Outcome: Change From Baseline in Immunoglobulin G (IgG) Subclasses up to 48 Weeks
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | Dimethyl Fumarate (BG00012)
Number analyzed (Participants) | 218
milligram per deciliter
  IgG Subclass 1: Baseline: number analyzed (Participants) | 189
  IgG Subclass 1: Baseline | 542.9 (152.87)
  IgG Subclass 1: Change at Week 4: number analyzed (Participants) | 169
  IgG Subclass 1: Change at Week 4 | -29.2 (68.22)
  IgG Subclass 1: Change at Week 8: number analyzed (Participants) | 170
  IgG Subclass 1: Change at Week 8 | -28.5 (71.46)
  IgG Subclass 1: Change at Week 12: number analyzed (Participants) | 182
  IgG Subclass 1: Change at Week 12 | -14.8 (79.07)
  IgG Subclass 1: Change at Week 24: number analyzed (Participants) | 170
  IgG Subclass 1: Change at Week 24 | -3.0 (78.80)
  IgG Subclass 1: Change at Week 36: number analyzed (Participants) | 163
  IgG Subclass 1: Change at Week 36 | -23.1 (61.73)
  IgG Subclass 1: Change at Week 48: number analyzed (Participants) | 166
  IgG Subclass 1: Change at Week 48 | -0.5 (102.41)
  IgG Subclass 2: Baseline: number analyzed (Participants) | 189
  IgG Subclass 2: Baseline | 350.7 (116.43)
  IgG Subclass 2: Change at Week 4: number analyzed (Participants) | 169
  IgG Subclass 2: Change at Week 4 | -22.7 (47.42)
  IgG Subclass 2: Change at Week 8: number analyzed (Participants) | 170
  IgG Subclass 2: Change at Week 8 | -26.5 (48.98)
  IgG Subclass 2: Change at Week 12: number analyzed (Participants) | 182
  IgG Subclass 2: Change at Week 12 | -18.9 (44.11)
  IgG Subclass 2: Change at Week 24: number analyzed (Participants) | 170
  IgG Subclass 2: Change at Week 24 | -5.5 (54.39)
  IgG Subclass 2: Change at Week 36: number analyzed (Participants) | 163
  IgG Subclass 2: Change at Week 36 | -22.4 (45.49)
  IgG Subclass 2: Change at Week 48: number analyzed (Participants) | 166
  IgG Subclass 2: Change at Week 48 | -21.5 (50.98)
  IgG Subclass 3: Baseline: number analyzed (Participants) | 189
  IgG Subclass 3: Baseline | 56.93 (26.860)
  IgG Subclass 3: Change at Week 4: number analyzed (Participants) | 169
  IgG Subclass 3: Change at Week 4 | -2.1 (8.56)
  IgG Subclass 3: Change at Week 8: number analyzed (Participants) | 170
  IgG Subclass 3: Change at Week 8 | -0.7 (12.36)
  IgG Subclass 3: Change at Week 12: number analyzed (Participants) | 182
  IgG Subclass 3: Change at Week 12 | -1.0 (15.48)
  IgG Subclass 3: Change at Week 24: number analyzed (Participants) | 170
  IgG Subclass 3: Change at Week 24 | -0.4 (11.31)
  IgG Subclass 3: Change at Week 36: number analyzed (Participants) | 163
  IgG Subclass 3: Change at Week 36 | 4.6 (19.09)
  IgG Subclass 3: Change at Week 48: number analyzed (Participants) | 166
  IgG Subclass 3: Change at Week 48 | 1.5 (12.55)
  IgG Subclass 4: Baseline: number analyzed (Participants) | 189
  IgG Subclass 4: Baseline | 30.35 (29.681)
  IgG Subclass 4: Change at Week 4: number analyzed (Participants) | 169
  IgG Subclass 4: Change at Week 4 | 1.24 (9.242)
  IgG Subclass 4: Change at Week 8: number analyzed (Participants) | 170
  IgG Subclass 4: Change at Week 8 | -0.38 (10.995)
  IgG Subclass 4: Change at Week 12: number analyzed (Participants) | 182
  IgG Subclass 4: Change at Week 12 | -0.12 (11.711)
  IgG Subclass 4: Change at Week 24: number analyzed (Participants) | 170
  IgG Subclass 4: Change at Week 24 | 1.08 (15.253)
  IgG Subclass 4: Change at Week 36: number analyzed (Participants) | 163
  IgG Subclass 4: Change at Week 36 | 1.28 (12.236)
  IgG Subclass 4: Change at Week 48: number analyzed (Participants) | 166
  IgG Subclass 4: Change at Week 48 | 3.26 (10.962)
  IgG Subclasses 1-4 Quant: Baseline: number analyzed (Participants) | 189
  IgG Subclasses 1-4 Quant: Baseline | 1029.9 (232.33)
  IgG Subclasses 1-4 Quant: Change at Week 4: number analyzed (Participants) | 169
  IgG Subclasses 1-4 Quant: Change at Week 4 | -54.6 (101.48)
  IgG Subclasses 1-4 Quant: Change at Week 8: number analyzed (Participants) | 170
  IgG Subclasses 1-4 Quant: Change at Week 8 | -41.9 (100.16)
  IgG Subclasses 1-4 Quant: Change at Week 12: number analyzed (Participants) | 181
  IgG Subclasses 1-4 Quant: Change at Week 12 | -28.5 (114.30)
  IgG Subclasses 1-4 Quant: Change at Week 24: number analyzed (Participants) | 170
  IgG Subclasses 1-4 Quant: Change at Week 24 | -55.7 (116.69)
  IgG Subclasses 1-4 Quant: Change at Week 36: number analyzed (Participants) | 164
  IgG Subclasses 1-4 Quant: Change at Week 36 | -70.3 (103.59)
  IgG Subclasses 1-4 Quant: Change at Week 48: number analyzed (Participants) | 167
  IgG Subclasses 1-4 Quant: Change at Week 48 | -65.1 (130.94)

ADVERSE EVENTS:
Time Frame: Up to 33 months
Description: The safety population was defined as all participants who received at least 1 dose of study treatment.
Arm/Group | Dimethyl Fumarate (BG00012)
All-Cause Mortality (participants affected / at risk) | 0/218
Serious Adverse Events (participants affected / at risk) | 26/218
Other Adverse Events (participants affected / at risk) | 160/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dimethyl Fumarate (BG00012) (N=218)
Acute myocardial infarction (Cardiac disorders) | 1
Iridocyclitis (Eye disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple sclerosis relapse (Nervous system disorders) | 16
Neurological decompensation (Nervous system disorders) | 1
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 1
Device malfunction (Product Issues) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dimethyl Fumarate (BG00012) (N=218)
Lymphopenia (Blood and lymphatic system disorders) | 13
Abdominal discomfort (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 22
Abdominal pain upper (Gastrointestinal disorders) | 22
Diarrhoea (Gastrointestinal disorders) | 28
Nausea (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 14
Fatigue (General disorders) | 27
Nasopharyngitis (Infections and infestations) | 33
Upper respiratory tract infection (Infections and infestations) | 28
Lymphocyte count decreased (Investigations) | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Headache (Nervous system disorders) | 16
Multiple sclerosis relapse (Nervous system disorders) | 41
Anxiety (Psychiatric disorders) | 13
Depression (Psychiatric disorders) | 12
Erythema (Skin and subcutaneous tissue disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 17
Flushing (Vascular disorders) | 100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT02525874/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT02525874/SAP_001.pdf